EudraCT Nº: 2016-002858-20

Version Number: 1.1 dated on 30/NOV/2017



# A PHASE II STUDY OF DURVALUMAB (MEDI4736) PLUS TREMELIMUMAB FOR THE TREATMENT OF PATIENTS WITH ADVANCED NEUROENDOCRINE NEOPLASMS OF GASTROENTEROPANCREATIC OR LUNG ORIGIN (THE DUNE TRIAL)

## STATISTICAL ANALYSIS PLAN (SAP)

| TRIAL FULL TITLE | A PHASE II STUDY OF DURVALUMAB (MEDI4736) PLUS TREMELIMUMAB FOR THE TREATMENT OF PATIENTS WITH ADVANCED NEUROENDOCRINE NEOPLASMS OF GASTROENTEROPANCREATIC OR LUNG ORIGIN (THE DUNE TRIAL) |
|---|---|
| EUDRACT NUMBER | 2016-002858-20DUNE |
| STUDY NUMBER | ESR 15-11561-DUNE |
| ISRCTN NUMBER | |
| INVESTIGATIONAL DRUG | DURVALUMAB (MEDI4736) AND TREMELIMUMAB |
| SAP VERSION | Version 1.1 |
| SAP VERSION DATE | 30/11/17 |
| TRIAL STATISTICIAN | |
| TRIAL CHIEF INVESTIGATOR | |
| SAP AUTHOR | |



Statistical Analysis Plan
Drug Substance DURVALUMAB/TREMELIMUMAB
Study Number ESR 15-11561-DUNE
EudraCT Nº: 2016-002858-20



## Version Number: 1.1 dated on 30/NOV/2017 1 GENERAL INFORMATION

#### TITLE

A phase II study of durvalumab (MEDI4736) plus tremelimumab for the treatment of patients with advanced neuroendocrine neoplasms of gastroenteropancreatic or lung origin (the DUNE trial).

#### STUDY DESIGN

Prospective, multi-center, open label, stratified, exploratory phase II study evaluating the efficacy and safety of durvalumab plus tremelimumab in different cohorts of patients with neuroendocrine neoplasms.

The study will include patients in four different cohorts:

- **Cohort 1**: Well-moderately differentiated lung neuroendocrine tumors (classically known as typical and atypical carcinoids) after progression to somatostatin analogs and one prior targeted therapy or chemotherapy.
- **Cohort 2**: G1/G2 (WHO grade 1 and 2) gastrointestinal neuroendocrine tumors after progression to somatostatin analogs and one prior targeted therapy.
- Cohort 3: G1/G2 (WHO grade 1 and 2) pancreatic neuroendocrine tumors after progression to standard therapies (chemotherapy, somatostatin analogs and target therapy), who have received between two and four prior lines of treatment.
- **Cohort 4**: Neuroendocrine neoplasms (WHO grade 3) of gastroenteropancreatic origin of unknown primary site (excluding lung primary tumors) after progression to first-line chemotherapy with a platinum based regimen.

#### **TREATMENT**

The treatment phase will include two stages for each cohort. The first stage will dose the first patient in each cohort in a safety run period for one cycle (4 weeks). If no unexpected side effects are observed in the first patient treated in each cohort during the safety run period, recruitment will continue up to 31 patients for cohorts 1 to 3, and 33 for cohort 4.

Subjects will be allocated in each primary tumour cohort to receive durvalumab 1500 mg Q4W for 12 months in patients plus tremelimumab 75 mg Q4W for up to 4 doses during the first 4 cycles of combined therapy. Cycles are defined by 4 weeks or 28 days. Subjects will undergo safety and efficacy assessment as defined per protocol.

#### **SPONSOR**

**GETNE** (Spanish Group of Neuroendocrine Tumors)

**Principal Investigators:** Dr. Jaume Capdevila

Statistical Analysis Plan
Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20




## **MONITORING ORGANISATION (CRO)**

| 1 | GEI | NERA | AL INFORMATION | 2 |
|---|-----|------|-------------------------------------------------------|----|
| 1 | ABI | BREV | IATIONS AND DEFINITIONS | 10 |
| 2 | INT | ROD | UCTION | 12 |
| | 2.1 | PRE | EFACE | 12 |
| | 2.2 | PUF | RPOSE OF THE ANALYSES | 12 |
| 3 | RES | SEAR | CH METHODS | 13 |
| | 3.1 | STL | JDY DESIGN | 13 |
| | 3.2 | STL | JDY OBJECTIVES | 13 |
| | 3.3 | STL | JDY POPULATION | 14 |
| | 3.3 | 3.1 | Sites | 14 |
| | 3.3 | 3.2 | Inclusion criteria | 14 |
| | 3.3 | 3.3 | Exclusion criteria | 16 |
| | 3.3 | 3.4 | Procedures for handling subjects incorrectly enrolled | 17 |
| | 3.4 | SCF | HEDULE OF STUDY PROCEDURES | 17 |
| | 3.5 | STU | JDY VARIABLES | 19 |
| | 3.5 | 5.1 | Schedule of study assessments | 21 |
| | 3.6 | SAN | MPLE SIZE | 24 |
| | 3.7 | DAT | TA ANALYSIS | 25 |
| | 3.7 | 7.1 | Analysis Sets | 25 |
| | 3.7 | 7.2 | Planned Analyses | 25 |
| | 3.7 | 7.3 | Planned Method of Analysis | 26 |
| | 3.7 | 7.4 | Data management and data cleaning | 26 |
| | 3.7 | 7.5 | Missing Data | 27 |
| | 3.7 | 7.6 | Interim Analyses | 27 |

Drug Substance DURVALUMAB/TREMELIMUMAB Study Number ESR 15-11561-DUNE

EudraCT Nº: 2016-002858-20

| | | | _ | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 10 | rc | in | 'n | Numb | or | 1 | • | 1 | date | bα | Oη | 30 | /NIO | 1/ | /20 | ٦1 | 7 |

Ve



| Ve | | mber: 1.1 dated on 30/NOV/2017 Neuroendocrinos | |
|---|---|---|---|
| | 3.7 | 5 | |
| | 3.7 | .8 SUMMARY OF STUDY DATA | 27 |
| | 3.8 | GENERAL CONSIDERATIONS | 27 |
| | 3.8.1 | Timing of Analyses | 27 |
| 1 | TAE | BLES, LISTING FIGURES | 29 |
| | 1.1 | STUDY POPULATION | 29 |
| | 1.1.1 | Recruited patients (sites/investigators) | 29 |
| | 1.1.2 | Analyzed patients | 29 |
| | 1.2 | DEMOGRAPHIC AND CLINICAL BASELINE CHARACTERISTICS | 32 |
| | 1.2.1 | Demographic and other baseline characteristics in cohort 1 | 38 |
| | 1.2.2 | Demographic and other baseline characteristics in cohort 2 | 44 |
| | 1.2.3 | Demographic and other baseline characteristics in cohort 3 | 50 |
| | 1.2.4 | Demographic and other baseline characteristics in cohort 4 | 56 |
| | 1.3 | STUDY MEDICATION | 62 |
| | 1.3.1 | Study medication in cohort 1 | 64 |
| | 1.3.2 | Study medication in cohort 2 | 65 |
| | 1.3.3 | Study medication in cohort 3 | 67 |
| | 1.3.4 | Study medication in cohort 4 | 69 |
| | 2 E | FFICACY ANALYSES | 71 |
| | 2.1 | PRIMARY EFFICACY ANALYSES | 71 |
| | 2.1.1 | Primary efficacy analyses in the Full Analysis Set | 71 |
| | 2.1.2 | Primary efficacy analyses in the Per Protocol Analysis Set | 73 |
| | 2.2 | SECONDARY EFFICACY ANALYSES | 75 |
| | 2.2.1 | Overall response rate (ORR) | 75 |
| | 2.2.2 | Response status at 6 and 12 months | 77 |
| | 2.2.3 | Progression Free Survival (PFS) | 80 |
| | 2.2.4 | Overall Survival (OS) | 88 |
| | 3 S | AFETY ANALYSES | 93 |
| | 3.1 | MOST FREQUENT TOXICITIES | 93 |
| | 3.2 | TOXICITIES GRADE≥3 | 94 |
| | 3.3 | EVERY TOXICITY | 96 |
| | 4 E | XPLORATORY ANALYSES | 97 |
| | 4.1<br>COHC | LOGISTIC REGRESSION: PREDICTOR FACTORS OF RESPONSE (CBR AT 9 MONTHS) IN E | |
| | 4.2 | COX REGRESSION: PREDICTOR FACTORS OF SURVIVAL IN EACH COHORT | 101 |

GETNE

Grupo Español de Tumores

Nauroendospinos

EudraCT Nº: 2016-002858-20 Version Number: 1.1 dated on 30/NOV/2017

| | | nber: 1.1 dated on 30/NOV/2017 | |
|---|-------|---------------------------------------------------------|-----|
| | 4.2.1 | Cox Regression: predictor factors of PFS in each cohort | 101 |
| | 4.2.2 | Cox Regression: predictor factors of OS in each cohort | 106 |
| 5 | GEN | IERAL CONSIDERATIONS | 110 |
| | 5.1 | TIMING OF ANALYSES | 110 |
| | 5.2 | REPORTING CONVENTIONS | 110 |
| | 5.3 | TECHNICAL DETAILS | 110 |
| 6 | RFF | FRENCES | 111 |

EudraCT Nº: 2016-002858-20




## **Tables**

| Table 1 Schedule of study assessments | 21 |
|---|---|
| Table 2 Recruited patients by Hospital | 29 |
| Table 3 Recruied patients and Analysis sets | 30 |
| Table 4 List of patients excluded from any of the analysis set | 30 |
| Table 5 Included/Excluded patients by Hospital | |
| Table 6 Patients allocated in each cohort by hospital | 31 |
| Table 7 Sociodemographic characteristics in overall | |
| Table 8 Vital signs in overall | 33 |
| Table 9 ECOG and PET in overall | 33 |
| Table 10 Tumor characteristics overall | 34 |
| Table 11 Baseline hematology laboratory test in overall | 34 |
| Table 12 Baseline clinical chemistry (serum or plasma) laboratory test in overall | 35 |
| Table 13 Baseline urinalysis test in overall | 35 |
| Table 14 Baseline TSH, fT3 and fT4 in overall | 36 |
| Table 15 Baseline coagulation in overall | 36 |
| Table 16 Hepatitis and HIV serologies in overall | 36 |
| Table 17 Disease-specific tumor markers and Anti PNS | 37 |
| Table 18 Concomitant medication | 37 |
| Table 19 Sociodemographic characteristics in overall in cohort 1 | 38 |
| Table 20 Vital signs in overall in cohort 1 | 38 |
| Table 21 ECOG and PET in overall in cohort 1 | 39 |
| Table 22 Tumor characteristics overall in cohort 1 | 39 |
| Table 23 Baseline hematology laboratory test in overall in cohort 1 | 40 |
| Table 24 Baseline clinical chemistry (serum or plasma) laboratory test in overall in cohort 1 | |
| Table 25 Baseline urinalysis test in overall in cohort 1 | 41 |
| Table 26 Baseline TSH, fT3 and fT4 in overall in cohort 1 | |
| Table 27 Baseline coagulation in overall in cohort 1 | 42 |
| Table 28 Hepatitis and HIV serologies in overall in cohort 1 | |
| Table 29 Disease-specific tumor markers and Anti PNS in cohort 1 | 42 |
| Table 30 Concomitant medication in cohort 1 | 43 |
| <b>0</b> 1 | 43 |
| Table 32 Vital signs in overall in cohort 2 | |
| Table 33 ECOG and PET in overall in cohort 2 | |
| Table 34 Tumor characteristics overall in cohort 2 | |
| Table 35 Baseline hematology laboratory test in overall in cohort 2 | |
| Table 36 Baseline clinical chemistry (serum or plasma) laboratory test in overall in cohort 2 | |
| Table 37 Baseline urinalysis test in overall in cohort 2 | |
| Table 38 Baseline TSH, fT3 and fT4 in overall in cohort 2 | |
| Table 39 Baseline coagulation in overall in cohort 2 | |
| Table 40 Hepatitis and HIV serologies in overall in cohort 2 | |
| Table 41 Disease-specific tumor markers and Anti PNS in cohort 2 | |
| Table 42 Concomitant medication in cohort 2 | |
| Table 43 Sociodemographic characteristics in overall in cohort 3 | 49 |

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20




| Table 44 Vital signs in overall in cohort 3 | 50 |
|---|---|
| Table 45 ECOG and PET in overall in cohort 3 | |
| Table 46 Tumor characteristics overall in cohort 3 | |
| Table 47 Baseline hematology laboratory test in overall in cohort 3 | 51 |
| Table 48 Baseline clinical chemistry (serum or plasma) laboratory test in overall in cohort 3 | |
| Table 49 Baseline urinalysis test in overall in cohort 3 | |
| Table 50 Baseline TSH, fT3 and fT4 in overall in cohort 3 | 53 |
| Table 51 Baseline coagulation in overall in cohort 3 | 53 |
| Table 52 Hepatitis and HIV serologies in overall in cohort 3 | 53 |
| Table 53 Disease-specific tumor markers and Anti PNS in cohort 3 | 54 |
| Table 54 Concomitant medication in cohort 3 | 54 |
| Table 55 Sociodemographic characteristics in overall in cohort 4 | 55 |
| Table 56 Vital signs in overall in cohort 4 | 55 |
| Table 57 ECOG and PET in overall in cohort 4 | |
| Table 58 Tumor characteristics overall in cohort 4 | |
| Table 59 Baseline hematology laboratory test in overall in cohort 4 | 57 |
| Table 60 Baseline clinical chemistry (serum or plasma) laboratory test in overall in cohort 4 | 57 |
| Table 61 Baseline urinalysis test in overall in cohort 4 | 58 |
| Table 62 Baseline TSH, fT3 and fT4 in overall in cohort 4 | |
| Table 63 Baseline coagulation in overall in cohort 4 | 58 |
| Table 64 Hepatitis and HIV serologies in overall in cohort 4 | 59 |
| Table 65 Disease-specific tumor markers and Anti PNS in cohort 4 | 59 |
| Table 66 Concomitant medication in cohort 4 | |
| Table 67 Clinical benefit rate (investigator assessment) at 9 months in the Full Analysis Set | 61 |
| Table 68 Overall survival rate at 9 months in the Full Analysis Set | |
| Table 69 Agreement in CBR by Cohen's kappa coefficient in the Full Analysis Set | 62 |
| Table 70 Clinical benefit rate (independent central radiology) at 9 months in the Full Analysis S | et62 |
| Table 71 Clinical benefit rate (investigator assessment) at 9 months in the Per Protocol Analysis | Set63 |
| Table 72 Overall survival rate at 9 months in the Per Protocol Analysis Set | 63 |
| Table 73 Agreement in CBR by Cohen's kappa coefficient in the Per Protocol Analysis Set | 63 |
| Table 74 Clinical benefit rate (independent central radiology) at 9 months in the Per Protocol | |
| Analysis Set | 64 |
| Table 75 ORR in the Full Analysis Set | 65 |
| Table 76 Duration of the response in the Full Analysis Set | |
| Table 77 ORR in the Per Protocol Analysis Set | |
| Table 78 Duration of the response in the Per Protocol Analysis Set | 67 |
| Table 79 Response status at 6 months in the Full Analysis Set | 67 |
| Table 80 Response status at 12 months in the Full Analysis Set | 68 |
| Table 81 Response status at 6 months in the Per Protocol Analysis Set | 68 |
| Table 82 Response status at 12 months in the Per Protocol Analysis Set | 69 |
| Table 83 Progression Free Survival in the Full Analysis Set | 70 |
| Table 84 Progression Free Survival in the Per-Protocol Analysis Set | 72 |
| Table 85 Overall Survival in the Full Analysis Set | 74 |
| Table 86 Overall Survival in the Per-Protocol Analysis Set | 76 |
| Table 87 Most frequent toxicities in overall | 78 |
| Table 88 Toxicities grade ≥3 during follow-up | 79 |
| Table 89 Every toxicity grade ≥3 in overall and by cohort | 79 |

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE

EudraCT Nº: 2016-002858-20




| version Number: 1.1 dated on 50/NOV/2017 | |
|---|---|
| Table 90 Details of every toxicity grade ≥3 by patient | 80 |
| Table 91 Patients with at least one toxicity during follow-up | 80 |
| Table 92 Every toxicity grade ≥3 in overall and by cohort | |
| Table 93 Univariate Logistic Regression for Response (CBR at 9 months) in cohort 1 (Full Analysi | S |
| Set) | |
| Table 94 Final multivariate Logistic Regression for Response (CBR at 9 months) in cohort 1 (Full | |
| Analysis Set) | |
| Table 95 Univariate Logistic Regression for Response (CBR at 9 months) in cohort 2 (Full Analysi | |
| Set) | |
| Table 96 Final multivariate Logistic Regression for Response (CBR at 9 months) in cohort 2 (Full | |
| Analysis Set) | |
| Table 97 Univariate Logistic Regression for Response (CBR at 9 months) in cohort 3 (Full Analysi | |
| Set) | |
| Table 98 Final multivariate Logistic Regression for Response (CBR at 9 months) in cohort 3 (Full | |
| Analysis Set) | |
| Table 99 Univariate Logistic Regression for Response (CBR at 9 months) in cohort 4 (Full Analysi | |
| Set) | |
| Table 100 Final multivariate Logistic Regression for Response (CBR at 9 months) in cohort 4 (Fu | |
| Analysis Set) | |
| Table 101 Univariate Cox Regression for PFS in cohort 1 (Full Analysis Set) | |
| Table 102 Final multivariate Cox Regression for PFS in cohort 1 (Full Analysis Set) | |
| Table 103 Univariate Cox Regression for PFS in cohort 2 (Full Analysis Set) | |
| Table 104 Final multivariate Cox Regression for PFS in cohort 2 (Full Analysis Set) | |
| Table 105 Univariate Cox Regression for PFS in cohort 3 (Full Analysis Set) | |
| Table 106 Final multivariate Cox Regression for PFS in cohort 3 (Full Analysis Set) | |
| Table 107 Univariate Cox Regression for PFS in cohort 4 (Full Analysis Set) | |
| Table 108 Final multivariate Cox Regression for PFS in cohort 4 (Full Analysis Set) | |
| Table 109 Univariate Cox Regression for OS in cohort 1 (Full Analysis Set) | |
| Table 110 Final multivariate Cox Regression for OS in cohort 1 (Full Analysis Set) | |
| Table 111 Univariate Cox Regression for OS in cohort 2 (Full Analysis Set) | |
| Table 112 Final multivariate Cox Regression for OS in cohort 2 (Full Analysis Set) | |
| Table 113 Univariate Cox Regression for OS in cohort 3 (Full Analysis Set) | |
| Table 114 Final multivariate Cox Regression for OS in cohort 3 (Full Analysis Set) | |
| Table 115 Univariate Cox Regression for OS in cohort 4 (Full Analysis Set) | |
| Table 116 Final multivariate Cox Regression for OS in cohort 4 (Full Analysis Set) | 93 |

EudraCT Nº: 2016-002858-20




## Figures:

| Figure 1. Progression Free Survival (Full Analysis Set) | 71 |
|-----------------------------------------------------------------|----|
| Figure 2. Progression Free Survival (Per-Protocol Analysis Set) | |
| Figure 3. Overall Survival (Full Analysis Set) | |
| Figure 4. Progression Free Survival (Per-Protocol Analysis Set) | |

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT №: 2016-002858-20




#### 1 ABBREVIATIONS AND DEFINITIONS

Abbreviation Explanation or special term

AchE Acetylcholine esterase

ADA Anti-drug antibody

AE Adverse event

AESI Adverse event of special interest
ALK Anaplastic lymphoma kinase
ALT Alanine aminotransferase

APF12 Proportion of patients alive and progression free at 12 months from

randomization

AST Aspartate aminotransferase

AUC Area under the curve

AUC0-28day Area under the plasma drug concentration-time curve from time zero to Day 28

post-dose

AUCss Area under the plasma drug concentration-time curve at steady state

BICR Blinded Independent Central Review

BoR Best objective response

BP Blood pressure

C Cycle

CD Cluster of differentiation
CI Confidence interval

CL Clearance

C<sub>max</sub> Maximum plasma concentration

C<sub>max,ss</sub> Maximum plasma concentration at steady state

CR Complete response
CSA Clinical study agreement
CSR Clinical study report
CT Computed tomography

CTCAE Common Terminology Criteria for Adverse Event CTLA-4 Cytotoxic T—lymphocyte-associated antigen 4

Ctrough,ss Trough concentration at steady state CXCL Chemokine (C-X-C motif) ligand

DoR Duration of response

EC Ethics Committee, synonymous to Institutional Review Board and Independent

**Ethics Committee** 

ECG Electrocardiogram

ECOG Eastern Cooperative Oncology Group

eCRF Electronic case report form
EdoR Expected duration of response
EGFR Epidermal growth factor receptor

EU European Union FAS Full analysis set

FDA Food and Drug Administration

GCP Good Clinical Practice
Gl Gastrointestinal

GMP Good Manufacturing Practice
hCG Human chorionic gonadotropin
HIV Human immunodeficiency virus

HR Hazard ratio

IB Investigator's Brochure

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20


ICF Informed consent form

ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee

IFN Interferon

IgE Immunoglobulin E
IgG Immunoglobulin G
IHC Immunohistochemistry

IL Interleukin

ILS Interstitial lung disease

IM Intramuscular

IMT Immunomodulatory therapy
IP Investigational product

irAE Immune-related adverse event
IRB Institutional Review Board

irRECIST Immune-related Response Evaluation Criteria in Solid Tumors

ITT Intent-to-Treat IV Intravenous

IVRS Interactive Voice Response System
IWRS Interactive Web Response System

mAb Monoclonal antibody

MDSC Myeloid-derived suppressor cell

MedDRA Medical Dictionary for Regulatory Activities
MHLW Minister of Health, Labor, and Welfare

miRNA Micro-ribonucleic acid
MRI Magnetic resonance imaging
NCI National Cancer Institute

NE Not evaluable

NSCLC Non-small-cell lung cancer
OAE Other significant adverse event

ORR Objective response rate

OS Overall survival
OSR Overall Survival Rate

PBMC Peripheral blood mononuclear cell

PD Progressive disease
PD-1 Programmed cell death 1

PD-L1 Programmed cell death ligand 1 PD-L2 Programmed cell death ligand 2

Pdx Pharmacodynamic(s)
PFS Progression-free survival
PFS2 Time to second progression
Pgx Pharmacogenetic research

PK Pharmacokinetic(s)
PR Partial response
q2w Every 2 weeks
q3w Every 3 weeks
q4w Every 4 weeks
q6w Every 6 weeks
q8w Every 8 weeks

QtcF QT interval corrected for heart rate using Fridericia's formula RECIST 1.1 Response Evaluation Criteria in Solid Tumors, version 1.1

RNA Ribonucleic acid



Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT №: 2016-002858-20

Version Number: 1.1 dated on 30/NOV/2017 RR Response rate

RT-QPCR Reverse transcription quantitative polymerase chain reaction

SAE Serious adverse event
SAP Statistical analysis plan
SAS Safety analysis set
SD Stable disease

SNP Single nucleotide polymorphism

SoC Standard of Care

sPD-L1 Soluble programmed cell death ligand 1

T<sub>3</sub> Triiodothyronine

T<sub>4</sub> Thyroxine

TSH Thyroid-stimulating hormone

ULN Upper limit of normal

UNK Unknown
US United States

WBDC Web-Based Data Capture WHO World Health Organization

#### 2 INTRODUCTION

#### 2.1 PREFACE

Neuroendocrine neoplasms constitute a heterogenic group of tumors derived from the Kultchitzky cells of the diffuse neuroendocrine system located in the gastrointestinal tract (origin of classical carcinoid tumors), pancreatic islet cells (origin of pancreatic endocrine tumors) and lung (origin of typical and atypical carcinoids). Advanced disease is common at diagnosis leading to limited options of curative strategies, so general prognosis is poor. Neuroendocrine neoplasms are considered rare diseases, however, taken all together into account and the natural history of well-differentiated tumors, their prevalence is increasing. Systemic treatment options have been limited for several years. However, in the last decade, the better knowledge of molecular biology of neuroendocrine neoplasms has increased the interest to develop targeted agents in this field, changing the scenario of possible therapies for advanced disease. Even though, treatment options are still limited.

Immune balance has always been related with neuroendocrine neoplasms. Prolonged stabilizations have often been described without treatment and initial immune modulators, such as interferon, have demonstrated antitumoral effects in these tumors. Recent advances in immunotherapy have permitted the development of new targeted agents with higher efficacy and lower toxicity that opens a new treatment option for patients with advanced neuroendocrine tumors.

#### 2.2 PURPOSE OF THE ANALYSES

These analyses will assess the efficacy and safety of durvalumab plus tremelimumab in different cohorts of patients with neuroendocrine neoplasms.



EudraCT Nº: 2016-002858-20




#### 3 RESEARCH METHODS

#### 3.1 STUDY DESIGN

Prospective, multi-center, open label, stratified, exploratory phase II study evaluating the efficacy and safety of durvalumab plus tremelimumab in different cohorts of patients with neuroendocrine neoplasms.

The study will include patients in four different cohorts:

- **Cohort 1**: Well-moderately differentiated lung neuroendocrine tumors (classically known as typical and atypical carcinoids) after progression to somatostatin analogs and one prior targeted therapy or chemotherapy.
- **Cohort 2**: G1/G2 (WHO grade 1 and 2) gastrointestinal neuroendocrine tumors after progression to somatostatin analogs and one prior targeted therapy.
- Cohort 3: G1/G2 (WHO grade 1 and 2) pancreatic neuroendocrine tumors after progression to standard therapies (chemotherapy, somatostatin analogs and target therapy), who have received between two and four prior lines of treatment.
- **Cohort 4**: Neuroendocrine neoplasms (WHO grade 3) of gastroenteropancreatic origin of unknown primary site (excluding lung primary tumors) after progression to first-line chemotherapy with a platinum based regimen.

#### 3.2 STUDY OBJECTIVES

#### **Primary Objectives:**

<u>Primary endpoint for cohorts 1, 2 and 3:</u> 9-months clinical benefit rate (CBR) by Response Evaluation Criteria In Solid Tumors (RECIST version 1.1).

Primary endpoint for cohort 4: 9-months overall survival rate.

#### Secondary Objective(s):

- Overall response rate (ORR) by irRECIST.
- To assess the duration of response according to irRECIST.
- To assess the median progression-free survival time (PFS) according to irRECIST.
- To assess the safety profile of durvalumab and tremelimumab in subjects with advanced neuroendocrine neoplasms.
- To assess the median overall survival (OS) time.
- To assess response status according to irRECIST at 6 and 12 months after start of study treatment.

#### **Exploratory Objective(s):**

To evaluate biochemical response (changes in CgA and NSE levels) and its association with

EudraCT Nº: 2016-002858-20


response rate and progression-free survival.



- To assess whether baseline tumor and blood biomarkers may be predictive of response to durvalumab and tremelimumab therapy.
- To explore additional hypotheses related to biomarkers and relationship to durvalumab and tremelimumab efficacy and/or toxicity and neuroendocrine tumors evolution that may arise from internal or external research activities.

#### 3.3 STUDY POPULATION

Patients with advanced/metastatic, histologically confirmed, grade 1/2 (G1/G2) of the 2010 WHO classification neuroendocrine tumors of the pancreas, gastrointestinal tract and lung origins and grade 3 (G3) of gastroenteropancreactic system or unknown primary site (excluding lung primaries) after progression to previous therapies.

#### 3.3.1 Sites

The selected study oncology sites in Spain were:

Hospital de Vall d'Hebron

Hospital

Hospital

Hospital

Hospital

Hospital

Hospital

Hospital

#### 3.3.2 **Inclusion criteria**

For inclusion in the study, patients should fulfill the following criteria:

- Written informed consent obtained from the subject prior to performing any protocolrelated procedures, including screening evaluations.
- 2. Age >18 years at time of study entry.
- 3. Subjects must have histologically confirmed diagnosis of one of the following advanced/metastatic neuroendocrine tumor types:
- Cohort 1: Well-moderately differentiated neuroendocrine tumors of the lung (Ki67<20% and mitotic count ≤20 mitoses x 10 HPF), also known as typical and atypical lung carcinoids, that have progressed to prior somatostatin analog therapy and/or one prior targeted therapy or chemotherapy (only one prior systemic therapy, with the exception of patients that have been treated with somatostatin analogues and other systemic treatment, when two prior treatments are allowed).
- Cohort 2: Well-moderately differentiated G1/G2 (WHO grade 1 and 2) gastrointestinal b) neuroendocrine tumors after progression to somatostatin analogs and one targeted therapy (prior targeted therapy could be everolimus or a multikinase inhibitor). Prior therapies with interferon alpha-2b or radionucleotide therapy are allowed.
- Cohort 3: Well-moderately differentiated neuroendocrine tumors G1/G2 (WHO grade 1 and 2) from pancreatic origin after progression to standard therapies (chemotherapy, somatostatin

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT №: 2016-002858-20




analogs and target therapy); patients must be treated with at least two prior systemic treatment lines and a maximum of four previous treatment lines.

- d) **Cohort 4:** Neuroendocrine neoplasms (WHO grade 3) of gastroenteropancreatic origin of unknown primary site (excluding lung primary tumors) after progression to first-line chemotherapy with a platinum based regimen.
- 4. For patients included in cohorts 1, 2 and 3: WHO Classification G1/G2 (Ki67<20% and mitotic count ≤20 mitoses x 10 HPF) lung typical and atypical carcinoids for cohort 1, gastrointestinal for cohort 2 (including stomach, small intestine and colorectal origins), pancreatic for cohort 3.
- 5. For patients included in cohort 4: WHO classification G3 (Ki67≥20% or mitotic count >20 mitoses x 10 HPF) gastroenteropancreatic neuroendocrine carcinomas (NEC) or liver metastases of G3 NEC of unknown primary site.
- 6. Subjects must have evidence of measurable disease meeting the following criteria:
- a) At least 1 lesion of  $\geq$  1.0 cm in the longest diameter for a non lymph node, or  $\geq$  1.5 cm in the short-axis diameter for a lymph node, which is serially measurable according to RECIST 1.1 (Appendix I) using computerized tomography/magnetic resonance imaging (CT/MRI). If there is only one target lesion and it is a non-lymph node, it should have a longest diameter of  $\geq$  1.5 cm.
- b) Lesions that have had external beam radiotherapy (EBRT) or loco-regional therapies such as radiofrequency (RF) ablation or liver embolization must show evidence of progressive disease based on RECIST 1.1 to be deemed a target lesion.
- c) Subjects must show evidence of disease progression by radiologic image techniques within 12 months (an additional month will be allowed to accommodate actual dates of performance of scans, i.e., within  $\leq$  13 months) prior to signing informed consent, according to RECIST 1.1 (Appendix I).
- 7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
- 8. Life expectancy of at least 12 weeks.
- 9. Adequate normal organ and marrow function as defined below:
- Haemoglobin ≥ 9.0 g/dL.
- Absolute neutrophil count (ANC)  $\geq 1.5 \times 10^9 / L$  (> 1500 per mm<sup>3</sup>).
- Platelet count  $\ge 100 \times 10^9 / L (>100,000 \text{ per mm}^3)$ .
- 1. Serum bilirubin  $\leq$  1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
- 2. AST (SGOT)/ALT (SGPT)  $\leq$  2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be  $\leq$  5x ULN.
- 3. Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

Males:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age)72 x serum creatinine (mg/dL)

Females:

Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85

72 x serum creatinine (mg/dL)

4. Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or

EudraCT Nº: 2016-002858-20


Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.



#### 3.3.3 **Exclusion criteria**

Subjects who meet any of the following criteria will be excluded from this study:

- Involvement in the planning and/or conduct of the study. 1.
- 2. Participation in another clinical study with an investigational product during the last 4 weeks.
- WHO Classification G3 neuroendocrine neoplasms of lung origin (oat cell/large cell lung 3. cancer).
- 4. Prior treatment with anti-PDL-1/anti-PD-1 or anti-CTL-4 therapy.
- 5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B (e.g., HBsAg reactive), hepatitis C (e.g., HCV RNA [qualitative] is detected) or known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
- 6. Known history of previous clinical diagnosis of tuberculosis.
- 7. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab or tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
- Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects 8. with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
- 9. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
- History of allogeneic organ transplant. 10.
- History of hypersensitivity to durvalumab, tremelimumab or any excipient. 11.
- Subjects having a diagnosis of immunodeficiency or are receiving systemic steroid therapy 12. or any other form of immunosuppressive therapy within 28 days prior to the first dose of trial treatment.
- 13. Knowledge of active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they have stable brain metastases [without evidence of progression by imaging confirmed [by magnetic resonance imaging (MRI) if MRI was used at prior imaging, or confirmed by computed tomography (CT) imaging if CT used at prior imaging] for at least four weeks prior to the first dose of trial treatment; also, any neurologic symptoms must have returned to baseline], have no evidence of new or enlarging brain metastases, and have not used steroids for brain metastases for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, as subjects with carcinomatous meningitis are excluded regardless of clinical stability.
- Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab or tremelimumab. Note: The killed virus vaccines used for seasonal influenza vaccines for injection are allowed; however intranasal influenza vaccines (e.g., FluMist®)



Statistical Analysis Plan Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20


are live attenuated vaccines, and are not allowed.



- 16. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1.
- Subjects who have received any anti-cancer treatment within 21 days or any investigational agent within 30 days prior to the first dose of study drug and should have recovered from any toxicity related to previous anti-cancer treatment. This does not apply to the use of somatostatin analogues for symptomatic therapy.
- Major surgery within 3 weeks prior to the first dose of study drug. 18.
- 19. Subjects having > 1+ proteinuria on urine dipstick testing will undergo 24h urine collection for quantitative assessment of proteinuria. Subjects with urine protein  $\geq 1$  g/24h will be ineligible.
- Significant cardiovascular impairment: history of congestive heart failure greater than New 20. York Heart Association (NYHA) Class II, unstable angina; myocardial infarction or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment.
- 21. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fredericia's Correction.
- Bleeding or thrombotic disorders or use of anticoagulants, such as warfarin, or similar agents requiring therapeutic international normalized ration (INR)monitoring. Treatment with low molecular weight heparin (LMWH) is allowed.
- 23. Active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug.
- 24. Active infection (any infection requiring treatment).
- Active malignancy (except for differentiated thyroid carcinoma, or definitively treated 25. melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix) within the past 24 months.
- 26. Known intolerance to any of the study drugs (or any of the excipients).
- 27. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ highly effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period.
- 28. Documented active alcohol or drug abuse.
- 29. Patients with a prior history of non-compliance with medical regimens.
- 30. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.

#### 3.3.4 Procedures for handling subjects incorrectly enrolled

Patients incorrectly enrolled in the trial will be considered as protocol desviations. If investigador considerer that the patient is obtaining benefit of the investigational treatment, patients could continue on therapy. They will not be considered for the primary endpoint of the trial, neither for efficacy nor biomarker secondary and exploratory analyses.

#### 3.4 SCHEDULE OF STUDY PROCEDURES

Before study entry, throughout the study, and following study drug discontinuation, various clinical and diagnostic laboratory evaluations are outlined. The purpose of obtaining these detailed measurements is to ensure adequate safety and tolerability assessments. Clinical evaluations and



EudraCT Nº: 2016-002858-20


laboratory studies may be repeated more frequently if clinically indicated.



#### Screening phase

Screening will occur between Day -28 and Day -1. The purpose of the screening period is to establish protocol eligibility. Informed consent will be obtained up to 4 weeks prior to Cycle 1 Day 1 and after the study has been fully explained to each subject and prior to the conduct of any screening procedures or assessments. The purpose of the baseline visit is to establish disease characteristics prior to allocation and treatment and to confirm protocol eligibility as specified in the inclusion/exclusion criteria. Results of baseline assessments must be obtained prior to the first dose of study drug (Cycle 1/Day 1). Baseline assessments may be performed on Day -1 or on Cycle 1/Day 1 prior to dosing. Clinical laboratory tests including pregnancy test (where applicable) can be performed within 72 hours of the first dose of study drug. Subjects who complete the baseline visit and continue to meet the criteria for inclusion/exclusion will begin the treatment phase of this study.

#### Treatment phase

The treatment phase will begin at the time of allocation of the first patient and will consist of the study treatment cycles. The treatment phase will end when the last patient discontinue the study drug. The treatment phase will include two stages for each cohort. The first stage will dose the first patient in each cohort in a safety run period for one cycle (4 weeks). If no unexpected side effects are observed in the first patient treated in each cohort during the safety run period, recruitment will continue up to 31 patients for cohorts 1 to 3, and 33 for cohort 4. Subjects will be allocated in each primary tumor cohort to receive durvalumab 1500 mg Q4W for 12 months in patients plus tremelimumab 75 mg Q4W for up to 4 doses during the first 4 cycles of combined therapy. Cycles are defined by 4 weeks or 28 days. Subjects will undergo safety and efficacy assessment as defined per protocol.

#### Follow-up phase

Patients will finish the treatment phase after the administration of 12 cycles of durvalumab or after disease progression during the treatment phase. For patients that complete all scheduled treatment, the follow-up phase will begin to determine survival endpoints. Tumor assessments will continue every 12 weeks and clinical appointments will start monthly during the first 3 months of follow-up and continue every 12 weeks until disease progression.

#### **End of Treatment**

#### End of treatment is defined as the last planned dosing visit within the 12-month dosing period.

For subjects who discontinue durvalumab or tremelimumab prior to 12 months, end of treatment is considered the last visit where the decision is made to discontinue treatment. All required procedures may be completed within ± 7 days of the end of treatment visit. Repeat disease assessment is not required if performed within 28 days prior to the end of treatment visit. Blood samples for biomarker analysis are collected. Assessments for subjects who have completed durvalumab and tremelimumab treatment and achieved disease control, or have discontinued durvalumab or tremelimumab due to toxicity in the absence of confirmed progressive disease are provided in APPENDIX 2 of the protocol.

Assessments for subjects who have discontinued durvalumab or tremelimumab treatment due to confirmed PD are presented in APPENDIX 3 of the protocol.

All subjects will be followed for survival until the end of the study regardless of further treatments,

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT №: 2016-002858-20

Version Number: 1.1 dated on 30/NOV/2017 or until the sponsor ends the study.



### 3.5 STUDY VARIABLES

#### Screening/Baseline variables:

- Hospital
- Informed Consent
- Eligibility criteria
- Allocated cohort
- Medical history and demographics (gender, date of birth and Race/ethnicity)
- Vital signs (temperature, respiratory rate, resting blood pressure, pulse), height and weight.
- ECOG performance status
- Concomitant medications
- 12-lead ECG (in triplicate [2-5 minutes apart])
- Record any Aes or SAEs (since ICF signature)
- Imaging by CT/MRI
- Review of octreoscan/PET (up to 6 months prior inclusion)
- Biomarkers analysis
- Archival tumor block or slides
- Clinical laboratory tests for:
- Hematology, Clinical chemistry, TSH, fT3 and fT4, Coagulation (PT, PTT, INR), Creatinine Clearance, Serum pregnancy test (for women of childbearing potential only), Hepatitis and VIH serologies, Urinalysis, Disease-specific tumor markers and Anti PNS.

#### **Tratment phase variables:**

#### Cycle 1/Day 1:

- Vital signs (temperature, respiratory rate, resting blood pressure, pulse) and weight.
- Administered study drug
- Concomitant medications
- Aes or SAEs

#### Cycle 1 to 3 / Day 15:

- Vital signs (temperature, respiratory rate, resting blood pressure, pulse) and weight.
- ECOG performance status
- Administered study drug
- Concomitant medications
- Aes or SAEs
- Biomarkers analysis
- Clinical laboratory tests for:
- Hematology, Clinical chemistry, TSH, fT3 and fT4, Coagulation (PT, PTT, INR), Creatinine Clearance, Serum pregnancy test (for women of childbearing potential only), Hepatitis and VIH serologies, Urinalysis, Disease-specific tumor markers and Anti PNS.

#### Cycle 2 to 12 /Day 1:

- Vital signs (temperature, respiratory rate, resting blood pressure, pulse) and weight.
- ECOG performance status
- Administered study drug (from C5D1 to C12D1 tremelimumab no longer administered, only

Statistical Analysis Plan Drug Substance DURVALUMAB/TREMELIMUMAB Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20


#### durvalumab).

- Biomarkers analysis
- Clinical laboratory tests for:
- Hematology, Clinical chemistry, TSH, fT3 and fT4, Coagulation (PT, PTT, INR), Creatinine Clearance ,Serum pregnancy test (for women of childbearing potential only),Hepatitis and VIH serologies, Urinalysis, Disease-specific tumor markers and Anti PNS.
- Concomitant medications
- Aes or SAEs
- Survival Data: Date and Status (alive/exitus)

#### Tumor assessments (CT/MRI)<sup>1</sup>

CT/MRI of chest/abdomen/pelvis and other areas of known disease at screening plus any areas of newly suspected disease should be performed every 8 weeks for the first 48 weeks and then every 12 weeks until confirmed PD (Date of assessment and status (PD or not PD)).



EudraCT Nº: 2016-002858-20




#### 3.5.1 Schedule of study assessments

#### Table 1 Schedule of study assessments

| Phase | Screenin | g Phase | | | | Treat | ment Phase | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Period | Screening a,b | Baseline <sup>a,b</sup> | | | | Study | / Treatment | | | | |
| Visit | V1<br>-28 to -2 | V2<br>Day -1 | V3<br>C1D1 | V4<br>C1D15 | V5<br>C2D1<br>(C1D28) | V6<br>C2D15 | V7<br>C3D1<br>(C2D28) | V8<br>C3D15 | V9<br>C4D1<br>(C3D28) | V10-V16<br>C5D1<br>C12D1 | Follow-up |
| Informed consent | Х | | | | | | | | | | |
| Inclusion/Exclusion | Х | Х | | | | | | | | | |
| Allocation | | Х | | | | | | | | | |
| Demographic Data | Х | | | | | | | | | | |
| ECOG PS <sup>C</sup> | Х | Х | | Х | Х | Х | Х | Х | Х | Х | Х |
| Prior Therapies for neuroendocrine neoplasms | х | | | | | | | | | | |
| Vitals signs <sup>d</sup> | X | | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Physical exam <sup>f</sup> | X | X <sup>e</sup> | | Х | Х | Х | Х | Х | Х | Х | Х |
| 12/lead ECG <sup>g</sup> | Х | | Only<br>when<br>clinically<br>indicated | | | | | | | | |
| Biochemistry and hematology <sup>h</sup> | х | X <sup>h</sup> | | Х | х | Х | Х | Х | Х | Х | Х |
| Hepatitis B and C; HIV | Х | | | | | | | | | | |

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE

EudraCT Nº: 2016-002858-20




| version Number: 1.1 dated on 30/ | NOV/2017 | 1 | | | 1 | iveuroendocrinos | | 1 | | 1 | 1 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Anti PNS antibody testing | Χ | | | | | | | | | | |
| Thyroid function test (TSH and fT3 and fT4) | Х | | | Х | Х | х | Х | Х | Х | х | Х |
| Urinalysis <sup>j</sup> | Х | | | Х | Х | Х | Х | Х | Х | Х | Х |
| Pregnancy test <sup>k</sup> | х | | Only<br>when<br>clinically<br>indicated | | | | | | | | |
| Durvalumab administration | | | Х | | Х | | Х | | Х | Х | |
| Tremelimumab administration | | | Х | | Х | | Х | | Х | | |
| Tumor assessments (CT/MRI) <sup>I</sup> | Х | | | | | | | s for the fir | | | reas of newly<br>ery 12 weeks |
| Octreoscan / PET/CT <sup>m</sup> | Х | | | | | | | | | | |
| Survival <sup>n</sup> | | | | | Х | | Х | | Х | Х | Х |
| Biomarkers <sup>o</sup> | | Х | | | Х | | | | | | |
| Archival tumor block or slides <sup>p</sup> | | х | | | | | | | | | |
| Concomitant medication | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | X |
| AEs/SAEs <sup>q</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | X |

AEs = adverse events, BP = blood pressure, CT = computerized tomography, ECG = electrocardiogram, ECOG = Eastern Cooperative Oncology Group, HR = heart rate, MRI = magnetic resonance imaging, PET = positron-emission tomography, RECIST = Response Evaluation Criteria In Solid Tumors, RR = respiratory rate, SAEs = serious adverse events, surg = surgical, 99m-Tc MDP = 99m-technetium-methylene diphosphonate, w/in = within.

a) 72 hours before Cycle 1 Day 1 (C1D1). The baseline assessment can be performed on C1D1, prior to treatment. Informed consent may be taken up to 4 weeks prior to C1D1.

EudraCT Nº: 2016-002858-20




- b) Efforts should be made to conduct study visits on the day scheduled (± 1 day). Clinical laboratory assessments may be conducted anytime within 72 hours prior to the scheduled visit.
- c) ECOG will be performed at the Screening and Baseline Visits and at every subsequent treatment visit thereafter. For ECOG see Appendix II of the protocol.
- d) Assessments will include vital signs (supine BP, HR, RR, and body temperature), weight, and height. Height will be measured at the Screening Visit only. Elevated BP (≥140/90 mmHg) should be confirmed by 3 measurements (at least 5 minutes apart). If systolic BP is ≥160 mmHg or diastolic BP ≥100 mmHg, BP should be confirmed by repeat measurements after an hour. Subjects will have their blood pressure and pulse measured before, during, and after the infusion at the following times (based on a 60-minute infusion):
- At the beginning of the infusion (at 0 minutes).
- At 30 minutes during the infusion (±5 minutes).
- At the end of the infusion (at 60 minutes ±5 minutes).
- In the 1 hour observation period post-infusion: 30 and 60 minutes after the infusion (ie, 90 and 120 minutes from the start of the infusion) (±5 minutes) for the first infusion only and then for subsequent infusions as clinically indicated.

If the infusion takes longer than 60 minutes, then blood pressure and pulse measurements should follow the principles as described above or more frequently if clinically indicated.

- e) Required if screening physical examination was performed > 7 days prior C1D1.
- f) A comprehensive physical examination (including a neurological examination) will be performed at the Screening or Baseline Visit, on each visit of the Treatment phase, and at the off-treatment assessment. A symptom-directed physical examination will be performed on Cycle 1/Day 1 and at any time during the study, as clinically indicated.
- g) Single 12-lead ECG. Subjects must be in the recumbent position for a period of 5 minutes prior to the ECG.
- h) Assessments scheduled may be performed within 72 hours prior to the visit. Assessments during follow up are made every 8-12 weeks, according to investigator's criteria.
- i) Free T3 and free T4 will only be measured if TSH is abnormal. They should also be measured if there is clinical suspicion of an adverse event related to the endocrine system. Assessments during follow up are made every 8-12 weeks, according to investigator's criteria.
- j) Assessments during follow up are made every 8-12 weeks, according to investigator's criteria.
- k) A serum or urine pregnancy test will be performed at the Screening Visit, at the Baseline Visit (or within 72 hours prior to the first dose of study medication).
- I) Screening tumor assessments using CT of the chest/abdomen/pelvis and other areas of known disease or newly suspected disease should be performed within 28 days prior to C1D1. Scans of the abdomen, pelvis and other areas of the body may be done with MRI instead of CT, but evaluation of the chest should be done with CT. CT scans should be performed with oral and iodinated IV contrast and MRI scans with IV gadolinium chelate unless there is a medical contraindication to contrast. If iodinated IV contrast is contraindicated, chest CT should be done without IV contrast.
- m) Somatostatin receptor schintigraphy (octreoscan) or PET-CT should be performed and/or available within the previous 6 months before C1D1.
- n) Survival data will be collected every 4 weeks until end of treatment phase is declared. All anticancer therapies will be collected. Survival data and other cancer treatments received will be collected every 6 months until close of the study database. The study sponsor may elect to discontinue survival follow-up.
- o) Collection of blood sample to obtain plasma, serum, or other components to be used for biomarker studies. Samples will be obtained at baseline, Cycle 2/Day 1, and at end-of-treatment visit.
- p) All subjects will have collection of most recent archived, tumor-biopsy sections for identification of predictive biomarkers.
- q) Throughout the study from the signature of Informed Consent. SAE irrespective of relationship to study treatment must be reported as soon as possible but not later than one business day. AEs and concomitant meds collected 28 days from last dose.

Statistical Analysis Plan
Drug Substance DURVALUMAB/TREMELIMUMAB
Study Number ESR 15-11561-DUNE
EudraCT Nº: 2016-002858-20




#### 3.6 SAMPLE SIZE

Sample size has been calculated using one-sample Superiority test (function OneSampleProportion. (NIS) of the Trial Size package of R software). According to previous knowledge, it is estimated that the reference value for the likelihood to be progression-free at 9 months is 30% and we expect an increase of 20% with a superiority margin of 10%. With a unilateral alpha level of 5% and 80% power, we estimate to include 28 patients per group, with an expected lost to follow-up rate of 10%, a final sample size in each 1, 2 and 3 cohort will include 31 patients.

For cohort 4, and according to previous knowledge, it is estimated that the reference proportion of patients being alive at 9 months is 13% and we expect an increase of 10% with a superiority margin of 5%. With a unilateral alpha level of 5% and 80% power, we estimate to include 30 patients per group, with an expected lost to follow-up rate of 10%, a final sample size will include 33 patients.

Summarizing, total sample size will include 126 patients: 31 patients for cohorts 1 to 3, and 33 for cohort 4.

EudraCT Nº: 2016-002858-20




#### 3.7 DATA ANALYSIS

#### 3.7.1 Analysis Sets

The analysis sets will be defined as follows:

- **Full Analysis Set** will include all allocated subjects. This will be primary analysis set for the efficacy endpoints.
- Per Protocol Analysis Set will include those subjects who were allocated and received at least one dose of the assigned study drug and had no major protocol deviations. The subjects will complete both baseline and at least one post-baseline tumor assessments (week 12).
- Safety Analysis Set will include all subjects who were allocated and received at least one dose of the study drug and had at least one post-baseline safety evaluation (week 12). This will be the analysis set for all safety evaluations.
- **Pharmacodynamic Analysis Set**: All the subjects who have received at least one dose of study drug and have evaluable pharmacodynamic data.

## 3.7.2 Planned Analyses

#### Demographic and other baseline characteristics

Demographic and other baseline characteristics will be summarized and listed. For continuous demographic/baseline variables including age, weight, and vital signs, results will be summarized and presented as n, number of not available data (NA), mean, standard deviation, median, and minimum and maximum values. For categorical variables such as race/ethnicity, the number and percentage of subjects will be used.

#### **Prior and concomitant medications**

Concomitant medications will be assigned an 11-digit code using the World Health Organization Drug Dictionary (WHO DD) drug codes. Concomitant medications will be further coded to the appropriate Anatomical-Therapeutic-Chemical (ATC) code indicating therapeutic classification. Prior and concomitant medications will be summarized and listed by drug and drug class.

#### **Efficacy Analyses**

All efficacy analyses will be based primarily on the Full Analysis Set and secondarily on the Per Protocol Analysis Set.

Data cut-off for the primary study analysis will happen following after the last patient included in the study has performed the first tumor evaluation (week 12 after first dose of study drug). The following tumor evaluations will take place every 12 weeks until documentation of disease progression or start of another anticancer therapy.

#### Analysis of primary efficacy variable

The analysis of clinical benefit rate and overall survival rate will be performed independently for each study cohort when the last patient included in the corresponding cohort of the study will arrived to 9 months after inclusion in the study or have progressed. The primary objective of the study will be based on the investigator assessment.

EudraCT Nº: 2016-002858-20




### 3.7.3 Planned Method of Analysis

Summary tables (descriptive statistics and frequency tables) will be provided for all baseline variables, efficacy variables, and safety variables, as appropriate. Continuous variables will be summarized with descriptive statistics (mean, standard deviation, range, and median). Ninety-five (95) percent confidence intervals (95% CI) may also be presented, as appropriate. Frequency counts and percentage of subjects within each category will be provided for categorical data.

The primary efficacy analysis will be performed using the binomial test procedure. Missing data will be treated using statistical multiple random imputation.

Concordance between investigator assessment and independent central radiology review will be analyzed using Cohen's Kappa. Although no significant differences are expected, a sensitivity analysis for the primary efficacy analysis will be performed using as response variable independent central radiology assessment.

Secondary endpoints will be summarized with descriptive statistics. Continuous variables will be summarized with n, mean, standard deviation, and range, frequency counts and percentage of subjects within each category will be provided for categorical data. Multivariate regression models will be used to study relations between explanatory variables and primary endpoint. Survival analysis will be performed to analyze PFS, Kaplan-Meier curves will be presented and possible comparisons will be tested using the log-rank test or the Cox proportional hazard model for multivariate analysis, hazard ratios (HR) and their 95% confidence interval (CI95%) will be provided. Patients with lost of follow-up or treatment discontinuation will be included in the final analysis of primary endpoint if they have at least one tumor evaluation and considered as censored data for survival endpoints.

R software version 3.2.1 will be used for all analysis.

#### Safety Analyses

Safety analyses will be based on the Safety Analysis Set. All safety analyses will be summarized separately by cohort. Adverse events and serious adverse events, laboratory test results, physical examination findings and vital signs, and their changes from baseline will be summarized using descriptive statistics. Abnormal values will be flagged.

## 3.7.4 Data management and data cleaning

Data was checked for inconsistencies, unexpected values and missing values. If identified, these values were fed back to the data contributor ( ), along with the patient identifier, for possible correction from source documents. Resubmitted, corrected, and/or transformed missing values were used to update the Data Base. If corrections could not be made, the inconsistencies and unexpected results are transformed to missing values.

*Missing dates:* In those cases that only the day was missing and month and year were known, in order to be able to use those dates for computing in the analysis, the date was rounded to day 15 of the month reported. Similarly, when month was not reported, the date was rounded to the sixth month of the year (June).

EudraCT Nº: 2016-002858-20




## 3.7.5 Missing Data

Assuming that the pattern of missingness in the primary endpoint variable (clinical benefit rate at 9 months) are missing at random (1), missing data will be treated using statistical multiple random imputation (2,3,4). Once date are collected, according to the missing data pattern observed, it should be considered if pre-specified methods are appropriate. A full reporting of all reasons for patient discontinuation should be given where possible, in order to identify the most important reasons that caused it. As suggested by the EMA (2), the seed of the pseudorandom number generator that will be used to randomly generate imputations for the missing values is prespecified ("55881234") to avoid bias being introduced by *post hoc* selection of the seed and therefore the random numbers to be imputed.

## 3.7.6 Interim Analyses

Not applicable

## 3.7.7 Data Monitoring

The sponsor's or representative (e.g., CRO's CRA) will maintain contact with the investigator and designated staff by telephone, and/or letter, and/or email between study visits. Monitoring visits to each investigational site will be conducted by the assigned CRA as described in the monitoring plan. The investigator (if regionally required, the heads of the medical institutions) will allow the CRA to inspect the clinical, laboratory, and pharmacy facilities to assure compliance with Good Clinical Practices and local regulatory requirements. The eCRFs and subject's corresponding original medical records (source documents) are to be fully available for review by the sponsor's representatives at regular intervals. These reviews verify adherence to the study protocol and data accuracy in accordance with federal regulations. All records at the investigational site, including source documents, are subject to inspection by the regulatory authorities and to review by the Ethical Committee.

#### 3.7.8 SUMMARY OF STUDY DATA

All continuous variables will be summarised using the following descriptive statistics: n (non-missing sample size), mean, standard deviation, median, maximum and minimum. The frequency and percentages (based on the non-missing sample size) of observed levels will be reported for all categorical measures. Frequency counts and percentage of subjects within each category will be provided for categorical data. Ninety-five (95) percent confidence intervals (95% CI) may also be presented, as appropriate. In general, all data will be listed, sorted by site, treatment and subject, and when appropriate by visit number within subject. All summary tables will be structured with a column for each cohort in the order (cohort 1, 2, 3 and 4) and will be annotated with the total population size relevant to that table/treatment, including any missing observations.

24 months

#### 3.8 GENERAL CONSIDERATIONS

## 3.8.1 Timing of Analyses

Recruitment period will be:

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT №: 2016-002858-20


Research Agreement executed: July 2016
 Projected IRB/IEC approval: Nov 2016
 First Subject In: Dec 2016
 50% Enrollment: Dec2017
 Last Subject In (100% enrollment): Dec 2018
 Last Subject Last Visit: Dec 2019
 Clinical Study Report April 2020

End of study is defined as Last Subject Last Visit.



EudraCT Nº: 2016-002858-20




## 1 TABLES, LISTING FIGURES

#### 1.1 STUDY POPULATION

## 1.1.1 Recruited patients (sites/investigators)

In this section, the number of recruited patients overall and by sites is listed.

#### Table 2 Recruited patients by Hospital

| | Hospital | n (%) |
|--------------|----------|-------|
| Hospital 1: | | |
| Hospital 2: | | |
| Hospital 3: | | |
| Hospital 4: | | |
| Hospital 5: | | |
| Hospital 6: | | |
| Hospital 7: | | |
| Hospital 8: | | |
| Hospital 9: | | |
| lospital 10: | | |
| Hospital 11: | | |
| Hospital 12: | | |
| Hospital 13: | | |
| Hospital 14: | | |
| Hospital 15: | | |
| Hospital 16: | | |
| Hospital 17: | | |
| Hospital 18: | | |
| Hospital 19: | | |
| Hospital 20: | | |
| Total | | |

## 1.1.2 Analyzed patients

If any patient is excluded from the study, it is listed in the table below, along with the reason for exclusion.

#### Table 3 Recruied patients and Analysis sets

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT №: 2016-002858-20




**Recruited patients** 100,0 Reason for exclusion - Reason1 - Reason 2 **Analysis Sets** Full Analysis Set: All allocated patients. Patients that fulfil Yes every inclusion criteria and none of the exclusion criteria, without any other reason for their exclusion No Per Protocol Analysis Set: Patients who were allocated and Yes received at least one dose of the assigned study drug and had no major protocol deviations. The subjects will complete both baseline and at least one post-baseline No tumor assessments (week 12). Safety Analysis Set: Patients who were allocated and Yes received at least one dose of the study drug and had at least one post-baseline safety evaluation (week 12). This No will be the analysis set for all safety evaluations. **Pharmacodynamic Analysis Set**: Patients who have Yes received at least one dose of study drug and have evaluable pharmacodynamic dats. No

In the following table, those patints excluded from any of the analysis sets will be listed along with the reasons for exclusion.

Table 4 List of patients excluded from any of the analysis set

| Number of patient | Cohort | Hospital | Analysis set | Reason for exclusion |
|-------------------|--------|----------|--------------|----------------------|

The number of patients included and excluded from each hospital will be reported.

#### Table 5 Included/Excluded patients by Hospital

| | Included | Excluded | Total |
|----------|----------|----------|-------|
| Hospital | n (%) | n (%) | n (%) |

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20




| Hospital 1 | |
|-------------|-----------|
| Hospital 2 | |
| Hospital 3 | |
| Hospital 4 | |
| Hospital 5 | |
| Hospital 6 | |
| Hospital 7 | |
| Hospital 8 | |
| Hospital 9 | |
| Hospital 10 | |
| Hospital 11 | |
| Hospital 12 | |
| Hospital 13 | |
| Hospital 14 | |
| Hospital 15 | |
| Hospital 16 | |
| Hospital 17 | |
| Hospital 18 | |
| Hospital 19 | |
| Hospital 20 | |
| Total | n (100.0) |

In the following table, the number of allocated patients in each one of the 4 cohorts by hospital will be shown.

Table 6 Patients allocated in each cohort by hospital

| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|------------|----------|----------|----------|----------|----------|
| Hospital | n (%) | n (%) | n (%) | n (%) | n (%) |
| Hospital 1 | | | | | n (100%) |
| Hospital 2 | | | | | n (100%) |
| Hospital 3 | | | | | n (100%) |
| Hospital 4 | | | | | n (100%) |
| Hospital 5 | | | | | n (100%) |
| Hospital 6 | | | | | n (100%) |
| Hospital 7 | | | | | n (100%) |
| Hospital 8 | | | | | n (100%) |
| Hospital 9 | | | | | n (100%) |

Height (cm)

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20




| Hospital 10 | n (100%) |
|-------------|----------|
| Hospital 11 | n (100%) |
| Hospital 12 | n (100%) |
| Hospital 13 | n (100%) |
| Hospital 14 | n (100%) |
| Hospital 15 | n (100%) |
| Hospital 16 | n (100%) |
| Hospital 17 | n (100%) |
| Hospital 18 | n (100%) |
| Hospital 19 | n (100%) |
| Hospital 20 | n (100%) |
| Total | n (100%) |

## 1.2 DEMOGRAPHIC AND CLINICAL BASELINE CHARACTERISTICS

For the descriptive analysis of the patients, the full analysis set is used (see section29).

#### Table 7 Sociodemographic characteristics in overall

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the<br>mean |
|---|---|---|---|---|---|
| Age (years) | | | | | |
| | | n | 9 | <sub>%</sub> 1 95 | % CI of the proportion |
| Gender | | | | | |
| Male | | | | | |
| Female | | | | | |
| UNK | | | | | |
| Race/ethnicity | | | | | |
| Caucasic | | | | | |
| Afro-american | | | | | |
| Others | | | | | |
| UNK | | | | | |
| <sup>1</sup> Calculated percent | age from | the total of patient | ts with available data | | |
| | | Table | 8 Vital signs in ov | erall | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the<br>mean |
| Weight (kg) | | | | | |

Statistical Analysis Plan Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20

2-10




| D | n | ЛI |
|---|----|----|
| В | I٧ | Ш |

| BMI | | | |
|---|---|---|---|
| Temperature | | | |
| Respiratory rate | | | |
| Systolic blood pressure | | | |
| Diastolic blood<br>pressure | | | |
| | Table 9 EC | OG in overall | |
| | n | <b>%</b> 1 | 95% CI of the proportion |
| ECOG | | | |
| 0 | | | |
| 1 | | | |
| 2 | | | |
| 3 | | | |
| 4 | | | |
| UNK | | | |
| <sup>1</sup> Calculated percentage from the | total of patients with av | ailable data | |
| | Table 10 Tumor cl | haracteristics overa | II |
| | n | %1 | 95% CI of the proportion |
| Histological type | | | |
| Well differentiated | | | |
| Moderately differentiated | | | |
| Poorly differentiated | | | |
| Ki-67 Index | | | |
| ≤2 | | | |
| 3-20 | | | |
| >20 | | | |
| Mitotic Index 10 CGA | | | |
| GEP-NETs | | | |
| <2 | | | |
| 2-20 | | | |
| >20 | | | |
| Lung/thymus | | | |
| <2 | | | |

Statistical Analysis Plan
Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20

>10




| Octreoscan/PET | | | | | | |
|---|---|---|---|---|---|---|
| Positive | | | | | | |
| Negative | | | | | | |
| Number or extranodal locations | | | | | | |
| 0 | | | | | | |
| 1 | | | | | | |
| 2 | | | | | | |
| 3 or more | | | | | | |
| UNK | | | | | | |
| <sup>1</sup> Calculated percent | age from i | the to | otal of patient | s with available | e data | |
| | | | | ical progression | | |
| | | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Time since radiological inclusion | PE to | | | | | |
| | Τα | able 1 | 12 Previous an | tineoplasic the | гару | |
| Name | n | | <b>%</b> 1 | | 95% CI of the p | roportion |
| Therapy 1 | | | | | | |
| Therapy 2 | | | | | | |
| Therapy 3 | | | | | | |
| Therapy 4 | | | | | | |
| Therapy 5 | | | | | | |
| Therapy 6 | | | | | | |
| <sup>1</sup> Calculated percentage | from the tot | tal of | patients with avo | ailable data | | |
| 7 | Table 13 B | est r | esponse to pre | evious antineop | lasic therapy | |
| | | n | <sub>%</sub> 1 | | 95% CI of the p | roportion |
| Complete response | | | | | | |
| Partial response | | | | | | |
| Stable Disease | | | | | | |
| Progression | | | | | | |
| UNK | | | | | | |
| Total | | | | | | |

 $<sup>^{</sup>f 1}$  Calculated percentage from the total of patients with available data

EudraCT Nº: 2016-002858-20




## Table 14 Baseline hematology laboratory test in overall

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|---|---|---|---|---|---|
| Basophils | | | | | |
| Eosinphils | | | | | |
| Hematocrit | | | | | |
| Hemoglobin | | | | | |
| Lymphocytes | | | | | |
| Mean corpuscular<br>hemoglobin | | | | | |
| Mean corpuscular hemoglobin concentration | | | | | |
| Mean corpuscular<br>volume | | | | | |
| Monocytes | | | | | |
| Neutrophils | | | | | |
| Platelet count | | | | | |
| Red blood cell count | | | | | |
| Total white cell count | | | | | |

## Table 15 Baseline clinical chemistry (serum or plasma) laboratory test in overall

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the<br>mean |
|---|---|---|---|---|---|
| Albumin | | | | | |
| Alkaline phosphatase | | | | | |
| Alanine aminotransferase | | | | | |
| Amylase | | | | | |
| Aspartate aminotransferase | | | | | |
| Bicarbonate | | | | | |
| Calcium | | | | | |
| Chloride | | | | | |
| Creatinine | | | | | |
| Clearance creatinine | | | | | |
| Gamma<br>glutamyltransferase | | | | | |

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20




mean

| Glucose | | | | | |
|---|---|---|---|---|---|
| Lactate<br>dehydrogenase | | | | | |
| Lipase | | | | | |
| Magnesium | | | | | |
| Potassium | | | | | |
| Sodium | | | | | |
| Total bilirubin | | | | | |
| Total protein | | | | | |
| Urea or blood urea<br>nitrogen, depending<br>on local practice | | | | | |
| Uric acid | | | | | |
| | | | seline urinalysis test | | 95% CI of the |
| | n | Mean (SD) | Median (IQR) | Min-Max | mean |
| Bilirubin | | | | | |
| Blood | | | | | |
| Glucose | | | | | |
| Ketones | | | | | |
| рН | | | | | |
| Protein | | | | | |
| Specific gravity | | | | | |
| Colour and appearance | | | | | |
| | | Table 17 Bas | eline TSH, fT3 and fT | 4 in overall | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the<br>mean |
| TSH | | | | | |
| fT3 | | | | | |
| fT4 | | | | | |
| | | Table 18 B | aseline coagulation | in overall | |
| | | n Mear | n (SD) Median (IQI | R) Min-Max | 95% CI of the |
Study Number ESR 15-11561-DI EudraCT Nº: 2016-002858-20


## GETNE Grupo Español de Tumores Neuroendocrinos

| Partial thromboplastin | Time |
|------------------------|------|
| (PTT) | |

**Neuron specific enolase** 

| <sup>1</sup> Calculated percentage from th | | | available data<br>c <b>tumor markers a</b> i | nd Anti PNS | |
|---|---|---|---|---|---|
| 1 Calculated percentage from th | e total | of nationts with a | available data | | |
| Negative | | | | | |
| Positive | | | | | |
| HIV | | | | | |
| Negative | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| Positive | | | | | |
| HBsAg | | | | | |
| Negative | | | | | |
| Positive | | | | | |
| Hepatitis HCV | | | | | |
| | | n | %1 | 95% CI | of the proportion |
| Т | able 1 | 9 Hepatitis an | nd HIV serologies in | n overall | |
| <sup>1</sup> Calculated percentage from | the to | tal of patients | with available data | | |
| UNK | | | | | |
| Negative | | | | | |
| Positive | | | | | |
| Anti PNS | | | | | |
| | | n | %1 | 95% CI of t | he proportion |
| International Normalized Ratio (INR) | | | | | |
| Prothrombin Time (PT) | | | | | |

Concomitant medications will be coded to the appropriate Anatomical-Therapeutic-Chemical (ATC) code indicating therapeutic classification. Prior and concomitant medications will be summarized and listed by drug and drug class.

EudraCT Nº: 2016-002858-20




| Concomitant medication Drug | | n | <b>%</b> 1 |
|-----------------------------|----------|---|------------|
| Drug class 1 | | | |
| | Drug 1.1 | | |
| | Drug 1.2 | | |
| | Drug 1 | | |
| Drug class 2 | | | |
| | Drug 2.1 | | |
| | Drug 2.2 | | |
| | Drug 2 | | |
| Drug class 3 | | | |
| | Drug 3.1 | | |
| | Drug 3.2 | | |
| | Drug 3 | | |

 $<sup>^{</sup>m 1}$  Calculated percentage from the total of patients with available data

## 1.2.1 Demographic and other baseline characteristics in cohort 1

For the descriptive analysis of the patients, the full analysis set is used (see section 29).

Table 22 Sociodemographic characteristics in overall in cohort 1

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the<br>mean |
|---|---|---|---|---|---|
| Age (years) | | | | | |
| | | n | 9 | <sub>%</sub> 1 95 | % CI of the proportion |
| Gender | | | | | |
| Male | | | | | |
| Female | | | | | |
| UNK | | | | | |
| Race/ethnicity | | | | | |
| Caucasic | | | | | |
| Afro-american | | | | | |
| Others | | | | | |
| UNK | | | | | |
| <sup>1</sup> Calculated percent | age from | the total of patient | s with available data | | |
| | | Table 23 Vit | al signs in overall | in cohort 1 | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the<br>mean |
| Weight (kg) | | | | | |

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20

<2




| version (valider: 1:1 dated on 30/100 1/2017 |
|----------------------------------------------|
| Llaight /am) |

| Height (cm) | • | | |
|---|---|---|---|
| ВМІ | | | |
| Temperature | | | |
| Respiratory rate | | | |
| Systolic blood pressure | | | |
| Diastolic blood<br>pressure | | | |
| | Table 24 ECOG | in overall in cohort 1 | |
| | n | <b>%</b> 1 | 95% CI of the proportion |
| ECOG | | | |
| 0 | | | |
| 1 | | | |
| 2 | | | |
| 3 | | | |
| 4 | | | |
| UNK | | | |
| $^{ m 1}$ Calculated percentage from the t | total of patients with | available data | |
| Tabl | le 25 Tumor chara | cteristics overall in coh | ort 1 |
| | n | <b>%</b> 1 | 95% CI of the proportion |
| Histological type | | | |
| Well differentiated | | | |
| Moderately differentiated | | | |
| Poorly differentiated | | | |
| Ki-67 Index | | | |
| ≤2 | | | |
| 3-20 | | | |
| >20 | | | |
| Mitotic Index 10 CGA | | | |
| GEP-NETs | | | |
| <2 | | | |
| 2-20 | | | |
| >20 | | | |
| Lung/thymus | | | |

Study Number ESR 15-11561-D EudraCT Nº: 2016-002858-20

UNK




| version Number. 1.1 dated | 1 011 30/ NO V/ 2017 | | | | | i veui delidoci illos |
|---|---|---|---|---|---|---|
| 2-10 | | | | | | |
| >10 | | | | | | |
| Octreoscan/PET | | | | | | |
| Positive | | | | | | |
| Negative | | | | | | |
| Number or extranoda | al | | | | | |
| locations | | | | | | |
| 0 | | | | | | |
| 1 | | | | | | |
| 2 | | | | | | |
| 3 or more | | | | | | |
| UNK | | | | | | |
| <sup>1</sup> Calculated percen | tage from the | e total of <sub>l</sub> | patient | ts with available | e data | |
| | | | | rogression to in | | rt 1 |
| | | | | | | 95% CI of the |
| | n | Mean | ı (SD) | Median (IQR) | Min-Max | mean |
| Time since radiologic inclusion | al PE to | | | | | |
| | Table 27 P | Previous a | ntineo <sub>l</sub> | plastic therapy | in cohort 1 | |
| Name | n | | <sub>%</sub> 1 | | 95% CI of the p | roportion |
| Therapy 1 | | | | | | |
| Therapy 2 | | | | | | |
| Therapy 3 | | | | | | |
| Therapy 4 | | | | | | |
| Therapy 5 | | | | | | |
| Therapy 6 | | | | | | |
| <sup>1</sup> Calculated percentage | e from the total | of patients | with av | ailable data | | |
| Table | 28 Best resp | onse to pr | evious | antineoplastic | therapy in coho | ort 1 |
| | n | | <sub>%</sub> 1 | <u> </u> | 95% CI of the p | proportion |
| Complete response | | | | | | |
| Partial response | | | | | | |
| Stable Disease | | | | | | |
| Progression | | | | | | |
| _ | | | | | | |

EudraCT Nº: 2016-002858-20






#### **Total**

### Table 29 Baseline hematology laboratory test in overall in cohort 1

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the<br>mean |
|---|---|---|---|---|---|
| Basophils | | | | | |
| Eosinphils | | | | | |
| Hematocrit | | | | | |
| Hemoglobin | | | | | |
| Lymphocytes | | | | | |
| Mean corpuscular hemoglobin | | | | | |
| Mean corpuscular hemoglobin concentration | | | | | |
| Mean corpuscular<br>volume | | | | | |
| Monocytes | | | | | |
| Neutrophils | | | | | |
| Platelet count | | | | | |
| Red blood cell count | | | | | |
| Total white cell count | | | | | |

#### Table 30 Baseline clinical chemistry (serum or plasma) laboratory test in overall in cohort 1

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|---|---|---|---|---|---|
| Albumin | | | | | |
| Alkaline phosphatase | | | | | |
| Alanine<br>aminotransferase | | | | | |
| Amylase | | | | | |
| Aspartate aminotransferase | | | | | |
| Bicarbonate | | | | | |
| Calcium | | | | | |
| Chloride | | | | | |
| Creatinine | | | | | |
| Clearance creatinine | | | | | |

 $<sup>\</sup>overline{\ ^{1}}$  Calculated percentage from the total of patients with available data

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE

EudraCT Nº: 2016-002858-20




| Gamma<br>glutamyltransferase | | | | | |
|---|---|---|---|---|---|
| Glucose | | | | | |
| Lactate<br>dehydrogenase | | | | | |
| Lipase | | | | | |
| Magnesium | | | | | |
| Potassium | | | | | |
| Sodium | | | | | |
| Total bilirubin | | | | | |
| Total protein | | | | | |
| Urea or blood urea nitrogen, depending on local practice | | | | | |
| Uric acid | | | | | |
| | Tab | le 31 Baseline | urinalysis test in ov | erall in cohort 1 | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the<br>mean |
| Bilirubin | | | | | |
| Blood | | | | | |
| Glucose | | | | | |
| Ketones | | | | | |
| рН | | | | | |
| Protein | | | | | |
| Specific gravity | | | | | |
| Colour and appearance | | | | | |
| | Table | 2 32 Baseline 1 | SH, fT3 and fT4 in o | verall in cohort 1 | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the<br>mean |
| TSH | | | | | |
| fT3 | | | | | |
| fT4 | | | | | |
| | Tal | ble 33 Baseline | e coagulation in ove | rall in cohort 1 | |
| | | | (OD) II (IO | | 95% CI of the |

Mean (SD)

n

Median (IQR)

Min-Max

mean

Grupo Español de Tumores

Neuroendocrinos

EudraCT Nº: 2016-002858-20




## Partial thromboplastin Time (PTT)

| Prothrombin Time (PT) | | | | | |
|---|---|---|---|---|---|
| International Normalized Ratio (INR) | | | | | |
| | | n | %1 | 95% CI of t | ne proportion |
| Anti PNS | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| UNK | | | | | |
| <sup>1</sup> Calculated percentage fro | om the to | tal of patients | with available data | | |
| Table | е 34 Нер | atitis and HIV | serologies in over | rall in cohort 1 | |
| | | n | <sub>%</sub> 1 | 95% CI | of the proportion |
| Hepatitis HCV | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| HBsAg | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| HBcAg | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| HIV | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| <sup>1</sup> Calculated percentage from | the total | of patients with a | vailable data | | |
| | | | or markers and An | ti PNS in cohor | t 1 |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Cg A | | | | | |
| Neuron specific enolase | | | | | |

Concomitant medications will be coded to the appropriate Anatomical-Therapeutic-Chemical (ATC) code indicating therapeutic classification. Prior and concomitant medications will be summarized and listed by drug and drug class.

EudraCT Nº: 2016-002858-20




| <b>Concomitant medication Drug</b> | | n | <b>%1</b> |
|------------------------------------|----------|---|-----------|
| Drug class 1 | | | |
| | Drug 1.1 | | |
| | Drug 1.2 | | |
| | Drug 1 | | |
| Drug class 2 | | | |
| | Drug 2.1 | | |
| | Drug 2.2 | | |
| | Drug 2 | | |
| Drug class 3 | | | |
| | Drug 3.1 | | |
| | Drug 3.2 | | |
| | Drug 3 | | |

 $<sup>^{</sup>f 1}$  Calculated percentage from the total of patients with available data

## 1.2.2 Demographic and other baseline characteristics in cohort 2

For the descriptive analysis of the patients, the full analysis set is used (see section 29).

Table 37 Sociodemographic characteristics in overall in cohort 2

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|---|---|---|---|---|---|
| Age (years) | | | | | |
| | | n | % | 1 95% ( | CI of the proportion |
| Gender | | | | | |
| Male | | | | | |
| Female | | | | | |
| UNK | | | | | |
| Race/ethnicity | | | | | |
| Caucasic | | | | | |
| Afro-american | | | | | |
| Others | | | | | |
| UNK | | | | | |
| <sup>1</sup> Calculated percenta | age from | the total of patient | s with available data | | |
| | | Table 38 Vit | tal signs in overall ir | n cohort 2 | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20 Version Number: 1.1 dated on

<2



| Version Number: 1.1 dated on 30/N | OV/2017 | | Neuroendocrinos |
|---|---|---|---|
| Height (cm) | | | |
| ВМІ | | | |
| Temperature | | | |
| Respiratory rate | | | |
| Systolic blood pressure | | | |
| Diastolic blood<br>pressure | | | |
| | Table 39 ECOG in | overall in cohort 2 | |
| | n | <sub>%</sub> 1 | 95% CI of the proportion |
| ECOG | | | |
| 0 | | | |
| 1 | | | |
| 2 | | | |
| 3 | | | |
| 4 | | | |
| UNK | | | |
| <sup>1</sup> Calculated percentage from th | ne total of patients with a | vailable data | |
| | ble 40 Tumor charact | | phort 2 |
| | n | <sub>%</sub> 1 | 95% CI of the proportion |
| Histological type | | | |
| Well differentiated | | | |
| Moderately differentiated | | | |
| Poorly differentiated | | | |
| Ki-67 Index | | | |
| ≤2 | | | |
| 3-20 | | | |
| >20 | | | |
| Mitotic Index 10 CGA | | | |
| GEP-NETs | | | |
| <2 | | | |
| 2-20 | | | |
| >20 | | | |
| Lung/thymus | | | |

Statistical Analysis Plan
Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20




| 2-10 | , , | | | | |
|---|---|---|---|---|---|
| >10 | | | | | |
| Octreoscan/PET | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| Number or extranodal locations | | | | | |
| 0 | | | | | |
| 1 | | | | | |
| 2 | | | | | |
| 3 or more | | | | | |
| UNK | | | | | |
| <sup>1</sup> Calculated percenta | ge from the t | otal of patient | s with available | e data | |
| | | | rogression to inc | | rt 2 |
| | | | | | 95% CI of the |
| | n | Mean (SD) | Median (IQR) | Min-Max | mean |
| Time since radiological I inclusion | PE to | | | | |
| | Table 42 Pre | vious antineor | olastic therapy i | n cohort 2 | |
| Name | Table 42 Pre | | plastic therapy i | | proportion |
| | | vious antineop<br>%1 | plastic therapy i | n cohort 2<br>95% CI of the p | roportion |
| Therapy 1 | | | plastic therapy i | | proportion |
| Therapy 1 Therapy 2 | | | olastic therapy i | | proportion |
| Therapy 1 Therapy 2 Therapy 3 | | | olastic therapy i | | proportion |
| Therapy 1 Therapy 2 Therapy 3 Therapy 4 | | | olastic therapy i | | proportion |
| Therapy 1 Therapy 2 Therapy 3 Therapy 4 Therapy 5 | | | olastic therapy i | | proportion |
| Therapy 1 Therapy 2 Therapy 3 Therapy 4 Therapy 5 Therapy 6 | n | <b>%1</b> | | | proportion |
| Therapy 1 Therapy 2 Therapy 3 Therapy 4 Therapy 5 Therapy 6 | n<br>rom the total of | %1 patients with ava | | 95% CI of the p | |
| Therapy 1 Therapy 2 Therapy 3 Therapy 4 Therapy 5 Therapy 6 | n<br>rom the total of | %1 patients with ava | ailable data<br>antineoplastic t | 95% CI of the p | ort 2 |
| Therapy 1 Therapy 2 Therapy 3 Therapy 4 Therapy 5 Therapy 6 | n<br>rom the total of<br>3 Best respon | %1<br>patients with avo | ailable data<br>antineoplastic t | 95% CI of the p | ort 2 |
| Therapy 1 Therapy 2 Therapy 3 Therapy 4 Therapy 5 Therapy 6 1 Calculated percentage fr Table 43 | n<br>rom the total of<br>3 Best respon | %1<br>patients with avo | ailable data<br>antineoplastic t | 95% CI of the p | ort 2 |
| Therapy 1 Therapy 2 Therapy 3 Therapy 4 Therapy 5 Therapy 6 1 Calculated percentage fr Table 43 Complete response | n<br>rom the total of<br>3 Best respon | %1<br>patients with avo | ailable data<br>antineoplastic t | 95% CI of the p | ort 2 |
| Therapy 1 Therapy 2 Therapy 3 Therapy 4 Therapy 5 Therapy 6 1 Calculated percentage fr Table 43 Complete response Partial response | n<br>rom the total of<br>3 Best respon | %1<br>patients with avo | ailable data<br>antineoplastic t | 95% CI of the p | ort 2 |
| Therapy 1 Therapy 2 Therapy 3 Therapy 4 Therapy 5 Therapy 6 1 Calculated percentage fr Table 43 Complete response Partial response Stable Disease | n<br>rom the total of<br>3 Best respon | %1<br>patients with avo | ailable data<br>antineoplastic t | 95% CI of the p | ort 2 |

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20




## $^{f 1}$ Calculated percentage from the total of patients with available data

#### Table 44 Baseline hematology laboratory test in overall in cohort 2

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the<br>mean |
|---|---|---|---|---|---|
| Basophils | | | | | |
| Eosinphils | | | | | |
| Hematocrit | | | | | |
| Hemoglobin | | | | | |
| Lymphocytes | | | | | |
| Mean corpuscular<br>hemoglobin | | | | | |
| Mean corpuscular<br>hemoglobin<br>concentration | | | | | |
| Mean corpuscular<br>volume | | | | | |
| Monocytes | | | | | |
| Neutrophils | | | | | |
| Platelet count | | | | | |
| Red blood cell count | | | | | |
| Total white cell count | | | | | |

#### Table 45 Baseline clinical chemistry (serum or plasma) laboratory test in overall in cohort 2

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|---|---|---|---|---|---|
| Albumin | | | | | |
| Alkaline phosphatase | | | | | |
| Alanine aminotransferase | | | | | |
| Amylase | | | | | |
| Aspartate aminotransferase | | | | | |
| Bicarbonate | | | | | |
| Calcium | | | | | |
| Chloride | | | | | |
| Creatinine | | | | | |
| Clearance creatinine | | | | | |
| Gamma | | | | | |

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20




| glutamyltransferase | | | | | |
|---|---|---|---|---|---|
| Glucose | | | | | |
| Lactate<br>dehydrogenase | | | | | |
| Lipase | | | | | |
| Magnesium | | | | | |
| Potassium | | | | | |
| Sodium | | | | | |
| Total bilirubin | | | | | |
| Total protein | | | | | |
| Urea or blood urea<br>nitrogen, depending<br>on local practice | | | | | |
| Uric acid | | | | | |
| | Tabl | le 46 Baselin | e urinalysis test i | n overall in cohort 2 | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the<br>mean |
| Bilirubin | | | | | |
| Blood | | | | | |
| Glucose | | | | | |
| Ketones | | | | | |
| рН | | | | | |
| Protein | | | | | |
| Specific gravity | | | | | |
| Colour and appearance | | | | | |
| | Table | 47 Baseline | TSH, fT3 and fT4 | in overall in cohort 2 | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| TSH | | | | | |
| fT3 | | | | | |
| fT4 | | | | | |
| | Tak | ole 48 Baselii | ne coagulation in | overall in cohort 2 | |
| | | n Mea | n (SD) Mediar | n (IQR) Min-Max | 95% CI of the mean |

Statistical Analysis Plan
Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT №: 2016-002858-20


# GETNE Grupo Español de Tumores Neuroendocrinos

## Partial thromboplastin Time (PTT)

Neuron specific enolase

| (· · · · ) | | | | | |
|---|---|---|---|---|---|
| Prothrombin Time (PT) | | | | | |
| International Normalized<br>Ratio (INR) | | | | | |
| | | n | %1 | 95% CI of t | he proportion |
| Anti PNS | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| UNK | | | | | |
| <sup>1</sup> Calculated percentage fi | rom the | total of patie | ents with available | e data | |
| Table | 49 Нер | atitis and HIV | serologies in over | rall in cohort 2 | |
| | | n | <b>%1</b> | 95% CI | of the proportion |
| Hepatitis HCV | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| HBsAg | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| HBcAg | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| HIV | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| <sup>1</sup> Calculated percentage from t | he total c | of patients with a | vailable data | | |
| Table 50 I | Disease | -specific tumo | or markers and An | ti PNS in cohor | t 2 |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Cg A | | | | | |

Concomitant medications will be coded to the appropriate Anatomical-Therapeutic-Chemical (ATC) code indicating therapeutic classification. Prior and concomitant medications will be summarized and listed by drug and drug class.

EudraCT Nº: 2016-002858-20




| Concomitant medication Drug | | n | <b>%</b> 1 |
|-----------------------------|----------|---|------------|
| rug class 1 | | | |
| | Drug 1.1 | | |
| | Drug 1.2 | | |
| | Drug 1 | | |
| Drug class 2 | | | |
| | Drug 2.1 | | |
| | Drug 2.2 | | |
| | Drug 2 | | |
| Drug class 3 | | | |
| | Drug 3.1 | | |
| | Drug 3.2 | | |
| | Drug 3 | | |

 $<sup>^{</sup>f 1}$  Calculated percentage from the total of patients with available data

## 1.2.3 Demographic and other baseline characteristics in cohort 3

For the descriptive analysis of the patients, the full analysis set is used (see section 29).

Table 52 Sociodemographic characteristics in overall in cohort 3

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|---|---|---|---|---|---|
| Age (years) | | | | | |
| | | n | % | 1 95% ( | CI of the proportion |
| Gender | | | | | |
| Male | | | | | |
| Female | | | | | |
| UNK | | | | | |
| Race/ethnicity | | | | | |
| Caucasic | | | | | |
| Afro-american | | | | | |
| Others | | | | | |
| UNK | | | | | |
| <sup>1</sup> Calculated percenta | age from | the total of patient | s with available data | | |
| | | Table 53 Vit | tal signs in overall ir | n cohort 3 | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20




| Height (cm) |
|-------------|
| BMI |

Temperature
Respiratory rate

Systolic blood

pressure

Diastolic blood

pressure

#### Table 54 ECOG in overall in cohort 3

| | n | <b>%1</b> | 95% CI of the proportion |
|------|---|-----------|--------------------------|
| ECOG | | | |
| 0 | | | |
| 1 | | | |
| 2 | | | |
| 3 | | | |
| 4 | | | |
| UNK | | | |

 $<sup>^{</sup> extstyle{1}}$  Calculated percentage from the total of patients with available data

#### Table 55 Tumor characteristics overall in cohort 3

| | n | <b>%</b> 1 | 95% CI of the proportion |
|---------------------------|---|------------|--------------------------|
| Histological type | | | |
| Well differentiated | | | |
| Moderately differentiated | | | |
| Poorly differentiated | | | |
| Ki-67 Index | | | |
| ≤2 | | | |
| 3-20 | | | |
| >20 | | | |
| Mitotic Index 10 CGA | | | |
| GEP-NETs | | | |
| <2 | | | |
| 2-20 | | | |
| >20 | | | |
| Lung/thymus | | | |
| <2 | | | |

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20




| 2-10 | | | | | | |
|---|---|---|---|---|---|---|
| >10 | | | | | | |
| Octreoscan/PET | | | | | | |
| Positive | | | | | | |
| Negative | | | | | | |
| Number or extranodal | | | | | | |
| locations | | | | | | |
| 0 | | | | | | |
| 1 | | | | | | |
| 2 | | | | | | |
| 3 or more | | | | | | |
| UNK | | | | | | |
| <sup>1</sup> Calculated percenta | age from t | the to | otal of patient | s with available | e data | |
| Table ! | 56 Time si | ince i | radiological pr | ogression to inc | clusion in coho | rt 3 |
| | | | | | | 95% CI of the |
| | | n | Mean (SD) | Median (IQR) | Min-Max | mean |
| Time since radiological P inclusion | PE to | | | | | |
| | Table 57 | 7 Pre | vious antineop | olastic therapy i | n cohort 3 | |
| Name | n | | % <sup>1</sup> | | 95% CI of the p | roportion |
| Therapy 1 | | | | | | |
| Therapy 2 | | | | | | |
| Therapy 3 | | | | | | |
| Therapy 4 | | | | | | |
| Therapy 5 | | | | | | |
| Therapy 6 | | | | | | |
| <sup>1</sup> Calculated percentage | from the | total | of patients with | h available data | | |
| Table 5 | 8 Best res | spons | se to previous | antineoplastic t | herapy in coho | ort 3 |
| | | n | %1 | | 95% CI of the p | roportion |
| Complete response | | | | | | |
| Partial response | | | | | | |
| Stable Disease | | | | | | |
| Stable Disease | | | | | | |

<sup>&</sup>lt;sup>1</sup>Calculated percentage from the total of patients with available data

EudraCT Nº: 2016-002858-20

Glucose




#### Table 59 Baseline hematology laboratory test in overall in cohort 3

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the<br>mean |
|---|---|---|---|---|---|
| Basophils | | | | | |
| Eosinphils | | | | | |
| Hematocrit | | | | | |
| Hemoglobin | | | | | |
| Lymphocytes | | | | | |
| Mean corpuscular hemoglobin | | | | | |
| Mean corpuscular hemoglobin concentration | | | | | |
| Mean corpuscular volume | | | | | |
| Monocytes | | | | | |
| Neutrophils | | | | | |
| Platelet count | | | | | |
| Red blood cell count | | | | | |
| Table 60 Baselin | e clin | nical chemistry ( | serum or plasma) lab | oratory test in ove | erall in cohort 3 |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Albumin | | | | | |
| Alkaline phosphatase | | | | | |
| Alanine aminotransferase | | | | | |
| Amylase | | | | | |
| Aspartate aminotransferase | | | | | |
| Bicarbonate | | | | | |
| Calcium | | | | | |
| Chloride | | | | | |
| Creatinine | | | | | |
| Clearance creatinine | | | | | |
| Gamma | | | | | |

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20




dehydrogenase Lipase

Magnesium

**Potassium** 

Sodium

**Total bilirubin** 

**Total protein** 

Urea or blood urea nitrogen, depending on local practice

**Uric acid** 

#### Table 61 Baseline urinalysis test in overall in cohort 3

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|---|---|---|---|---|---|
| Bilirubin | | | | | |
| Blood | | | | | |
| Glucose | | | | | |
| Ketones | | | | | |
| рH | | | | | |
| Protein | | | | | |
| Specific gravity | | | | | |
| Colour and appearance | | | | | |

#### Table 62 Baseline TSH, fT3 and fT4 in overall in cohort 3

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the<br>mean |
|-----|---|-----------|--------------|---------|-----------------------|
| TSH | | | | | |
| fT3 | | | | | |
| fT4 | | | | | |

#### Table 63 Baseline coagulation in overall in cohort 3

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the<br>mean |
|---|---|---|---|---|---|
| Partial thromboplastin Time (PTT) | | | | | |
| Prothrombin Time (PT) | | | | | |



Statistical Analysis Plan Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20




| | | n | 0/4 | | |
|---|---|---|---|---|---|
| | | n | %1 | 95% CI of tl | ne proportion |
| Anti PNS | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| UNK | | | | | |
| <sup>1</sup> Calculated percentage from | the to | tal of patients | with available data | 1 | |
| Table 6 | 64 Нер | atitis and HIV | serologies in over | rall in cohort 3 | |
| | | n | <b>%</b> 1 | 95% CI | of the proportion |
| Hepatitis HCV | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| HBsAg | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| HBcAg | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| HIV | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| $^{ m 1}$ Calculated percentage from th | ne total o | of patients with a | vailable data | | |
| Table 65 D | Disease | -specific tumo | or markers and An | nti PNS in cohor | t 3 |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Cg A | | | | | |
| Neuron specific enolase | | | | | |

and listed by drug and drug class.

#### Table 66 Concomitant medication in cohort 3

| Concomitant medication Drug n %1 |
|----------------------------------|
|----------------------------------|

EudraCT Nº: 2016-002858-20




#### Drug class 1

| | Drug 1.1 |
|--------------|----------|
| | Drug 1.2 |
| | Drug 1 |
| Drug class 2 | |
| | Drug 2.1 |
| | Drug 2.2 |
| | Drug 2 |
| Drug class 3 | |
| | Drug 3.1 |
| | Drug 3.2 |
| | Drug 3 |

 $<sup>^{</sup>f 1}$  Calculated percentage from the total of patients with available data

## 1.2.4 Demographic and other baseline characteristics in cohort 4

For the descriptive analysis of the patients, the full analysis set is used (see section 29).

Table 67 Sociodemographic characteristics in overall in cohort 4

| | | • | • | | |
|---|---|---|---|---|---|
| | n | Mean (SD) | Median (IQR) | Min-Ma | 95% CI of the<br>mean |
| Age (years) | | | | | |
| | | n | | <sub>%</sub> 1 | 95% CI of the proportion |
| Gender | | | | | |
| Male | | | | | |
| Female | | | | | |
| UNK | | | | | |
| Race/ethnicity | | | | | |
| Caucasic | | | | | |
| Afro-american | | | | | |
| Others | | | | | |
| UNK | | | | | |
| <sup>1</sup> Calculated percenta | ige from | the total of patient | s with available data | 3 | |
| | | Table 68 Vit | tal signs in overa | ll in cohort 4 | |
| | n | Mean (SD) | Median (IQR) | Min-Ma | 95% CI of the<br>mean |
| Weight (kg) | | | | | |
| Height (cm) | | | | | |

EudraCT Nº: 2016-002858-20




| п | n | л | |
|---|----|----|---|
| В | I١ | /1 | ı |

| Temperature |
|-----------------------------|
| Respiratory rate |
| Systolic blood<br>pressure |
| Diastolic blood<br>pressure |

#### Table 69 ECOG in overall in cohort 4

| | n | <sub>%</sub> 1 | 95% CI of the proportion |
|------|---|----------------|--------------------------|
| ECOG | | | |
| 0 | | | |
| 1 | | | |
| 2 | | | |
| 3 | | | |
| 4 | | | |
| UNK | | | |

 $<sup>^{</sup> extstyle{1}}$  Calculated percentage from the total of patients with available data

#### Table 70 Tumor characteristics overall in cohort 4

| | n | <b>%1</b> | 95% CI of the proportion |
|---------------------------|---|-----------|--------------------------|
| Histological type | | | |
| Well differentiated | | | |
| Moderately differentiated | | | |
| Poorly differentiated | | | |
| Ki-67 Index | | | |
| ≤2 | | | |
| 3-20 | | | |
| >20 | | | |
| Mitotic Index 10 CGA | | | |
| GEP-NETs | | | |
| <2 | | | |
| 2-20 | | | |
| >20 | | | |
| Lung/thymus | | | |
| <2 | | | |
| 2-10 | | | |

Statistical Analysis Plan
Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20




| >10 | | | | | |
|---|---|---|---|---|---|
| Octreoscan/PET | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| Number or extranoda | al | | | | |
| locations | | | | | |
| 0 | | | | | |
| 1 | | | | | |
| 2 | | | | | |
| 3 or more | | | | | |
| UNK | | | | | |
| <sup>1</sup> Calculated percen | tage from the | total of patien | ts with available | data | |
| | | | rogression to inc | | rt 4 |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Time since radiologica inclusion | al PE to | | | | |
| | Table 72 P | revious antineo | plastic therapy ii | n cohort 4 | |
| Name | n | <b>%1</b> | | 95% CI of the p | proportion |
| Therapy 1 | | | | | |
| Therapy 2 | | | | | |
| Therapy 3 | | | | | |
| Therapy 4 | | | | | |
| Therapy 5 | | | | | |

#### Table 73 Best response to previous antineoplastic therapy in cohort 4

<sup>1</sup>Calculated percentage from the total of patients with available data

| | n | <b>%1</b> | 95% CI of the proportion |
|-------------------|---|-----------|--------------------------|
| Complete response | | | |
| Partial response | | | |
| Stable Disease | | | |
| Progression | | | |
| UNK | | | |

EudraCT Nº: 2016-002858-20






<sup>1</sup>Calculated percentage from the total of patients with available data

#### Table 74 Baseline hematology laboratory test in overall in cohort 4

| | | | | | 95% CI of the |
|---|---|---|---|---|---|
| | n | Mean (SD) | Median (IQR) | Min-Max | mean |
| Basophils | | | | | |
| Eosinphils | | | | | |
| Hematocrit | | | | | |
| Hemoglobin | | | | | |
| Lymphocytes | | | | | |
| Mean corpuscular hemoglobin | | | | | |
| Mean corpuscular hemoglobin concentration | | | | | |
| Mean corpuscular<br>volume | | | | | |
| Monocytes | | | | | |
| Neutrophils | | | | | |
| Platelet count | | | | | |
| Red blood cell count | | | | | |
| Total white cell count | | | | | |

#### Table 75 Baseline clinical chemistry (serum or plasma) laboratory test in overall in cohort 4

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|---|---|---|---|---|---|
| Albumin | | | | | |
| Alkaline phosphatase | | | | | |
| Alanine aminotransferase | | | | | |
| Amylase | | | | | |
| Aspartate aminotransferase | | | | | |
| Bicarbonate | | | | | |
| Calcium | | | | | |
| Chloride | | | | | |
| Creatinine | | | | | |

EudraCT Nº: 2016-002858-20




| Clearance creatinine | | | | | |
|---|---|---|---|---|---|
| Gamma<br>glutamyltransferase | | | | | |
| Glucose | | | | | |
| Lactate<br>dehydrogenase | | | | | |
| Lipase | | | | | |
| Magnesium | | | | | |
| Potassium | | | | | |
| Sodium | | | | | |
| Total bilirubin | | | | | |
| Total protein | | | | | |
| Urea or blood urea nitrogen, depending on local practice | | | | | |
| Uric acid | | | | | |
| | Tabi | le 76 Baseline | urinalysis test in o | verall in cohort 4 | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Bilirubin | | | | | |
| Blood | | | | | |
| Glucose | | | | | |
| Ketones | | | | | |
| рН | | | | | |
| Protein | | | | | |
| Specific gravity | | | | | |
| Colour and appearance | | | | | |
| | Table | 77 Baseline T | SH, fT3 and fT4 in o | overall in cohort 4 | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| TSH | | | | | |
| fT3 | | | | | |
| fT4 | | | | | |

Study Number ESR 15-11561-DU EudraCT Nº: 2016-002858-20




| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|---|---|---|---|---|---|
| Partial thromboplastin Time (PTT) | | | | | |
| Prothrombin Time (PT) | | | | | |
| International Normalized<br>Ratio (INR) | | | | | |
| | | n | %1 | 95% CI of t | he proportion |
| Anti PNS | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| UNK | | | | | |
| <sup>1</sup> Calculated percentage from | the to | tal of patients | with available data | 1 | |
| Table 7 | 79 Нер | atitis and HIV | serologies in ove | rall in cohort 4 | |
| | | n | <b>%</b> 1 | 95% CI | of the proportion |
| Hepatitis HCV | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| HBsAg | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| HBcAg | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| HIV | | | | | |
| Positive | | | | | |
| Negative | | | | | |
| $^{ m 1}$ Calculated percentage from th | e total | of patients with a | available data | | |
| Table 80 D | Disease | e-specific tumo | or markers and An | nti PNS in cohor | t 4 |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Cg A | | | | | |
| Neuron specific enolase | | | | | |

Concomitant medications will be coded to the appropriate Anatomical-Therapeutic-Chemical (ATC) code indicating therapeutic classification. Prior and concomitant medications will be summarized

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20

Version Number: 1.1 dated on 30/NOV/2017 and listed by drug and drug class.



#### Table 81 Concomitant medication in cohort 4

| Concomitant medication Drug | | n | <b>%1</b> |
|-----------------------------|----------|---|-----------|
| Drug class 1 | | | |
| | Drug 1.1 | | |
| | Drug 1.2 | | |
| | Drug 1 | | |
| Drug class 2 | | | |
| | Drug 2.1 | | |
| | Drug 2.2 | | |
| | Drug 2 | | |
| Drug class 3 | | | |
| | Drug 3.1 | | |
| | Drug 3.2 | | |
| | Drug 3 | | |

 $<sup>^{</sup>f 1}$  Calculated percentage from the total of patients with available data

### 1.3 STUDY MEDICATION

For the descriptive analysis of the patients, the full analysis set is used (see section 29).

Table 82 Adherence to Durvalumab

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|---|---|---|---|---|---|
| Cycles received | | | | | |
| 12 Cycles received | | n | <b>%</b> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| Cycles received | | n | <b>%</b> 1 | 95% CI o | f the proportion |
| 0 | | | | | |
| 1 | | | | | |
| 2 | | | | | |
| 3 | | | | | |
| 4 | | | | | |
| 5 | | | | | |
| 6 | | | | | |
| 7 | | | | | |
| 8 | | | | | |

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20



| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|---|---|---|---|---|---|
| | | Table 83 A | dherence to Treme | limumab | |
| <sup>1</sup> Calculated percenta | ge from t | he total of patien | ts with available data | | |
| Cycles omitted | | | | | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| No | | | | | |
| Yes | | | | | |
| Cycles omitted | | n | <b>%1</b> | 95% CI o | f the proportion |
| Cycles delayed | | | | | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| No | | | | | |
| Yes | | | | | |
| Cycles delayed | | n | <b>%</b> 1 | 95% CI o | f the proportion |
| 12 | | | | | |
| 11 | | | | | |
| 10 | | | | | |
| 9 | | | | | |
| Version Number: 1.1 dat | | NOV/2017 | | | Neuroendocrinos |

| | 11 | iviean (SD) | wedian (IQK) | IVIIII-IVIAX | 95% Ci oi the mean |
|---|---|---|---|---|---|
| Cycles received | | | | | |
| 4 Cycles received | | n | <sub>%</sub> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| Cycles received | | n | <b>%</b> 1 | 95% CI o | f the proportion |
| 0 | | | | | |
| 1 | | | | | |
| 2 | | | | | |
| 3 | | | | | |
| 4 | | | | | |
| Cycles delayed | | n | <b>%</b> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Cycles delayed | | | | | |
| Cycles omitted | | n | <b>%</b> 1 | 95% CI of the proportion | |
| Yes | | | | | |
| No | | | | | |

Study Number ESR 15-11561-DI EudraCT Nº: 2016-002858-20




| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|----------------|---|-----------|--------------|---------|--------------------|
| Cycles omitted | | | | | |

 $<sup>\</sup>overline{\phantom{a}^1}$  Calculated percentage from the total of patients with available data

## 1.3.1 Study medication in cohort 1

For the descriptive analysis of the patients, the full analysis set is used (see section 29).

#### Table 84 Adherence to Durvalumab in cohort 1

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|---|---|---|---|---|---|
| Cycles received | | | | | |
| 12 Cycles received | | n | <b>%</b> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| Cycles received | | n | <b>%1</b> | 95% CI o | f the proportion |
| 0 | | | | | |
| 1 | | | | | |
| 2 | | | | | |
| 3 | | | | | |
| 4 | | | | | |
| 5 | | | | | |
| 6 | | | | | |
| 7 | | | | | |
| 8 | | | | | |
| 9 | | | | | |
| 10 | | | | | |
| 11 | | | | | |
| 12 | | | | | |
| Cycles delayed | | n | <b>%1</b> | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Cycles delayed | | | | | |
| Cycles omitted | | n | <b>%</b> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |

Study Number ESR 15-11561-DUNE EudraCT №: 2016-002858-20




| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|----------------|---|-----------|--------------|---------|--------------------|
| Cycles omitted | | | | | |

 $<sup>\</sup>overline{\phantom{a}^1}$  Calculated percentage from the total of patients with available data

#### Table 85 Adherence to Tremelimumab in cohort 1

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|---|---|---|---|---|---|
| Cycles received | | | | | |
| 4 Cycles received | | n | <sub>%</sub> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| Cycles received | | n | <b>%</b> 1 | 95% CI o | f the proportion |
| 0 | | | | | |
| 1 | | | | | |
| 2 | | | | | |
| 3 | | | | | |
| 4 | | | | | |
| Cycles delayed | | n | <b>%</b> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Cycles delayed | | | | | |
| Cycles omitted | | n | <sub>%</sub> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Cycles omitted | | | | | |

 $<sup>^{\,1}</sup>$  Calculated percentage from the total of patients with available data

## 1.3.2 Study medication in cohort 2

For the descriptive analysis of the patients, the full analysis set is used (see section 29).

#### Table 86 Adherence to Durvalumab in cohort 2

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|---|---|---|---|---|---|
| Cycles received | | | | | |
| 12 Cycles received | | n | <b>%</b> 1 | 95% CI of the proportion | |
| Yes | | | | | |
| No | | | | | |

Statistical Analysis Plan
Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20

2




| Cycles received | | n | <b>%</b> 1 | 95% CI o | f the proportion |
|---|---|---|---|---|---|
| 0 | | | | | |
| 1 | | | | | |
| 2 | | | | | |
| 3 | | | | | |
| 4 | | | | | |
| 5 | | | | | |
| 6 | | | | | |
| 7 | | | | | |
| 8 | | | | | |
| 9 | | | | | |
| 10 | | | | | |
| 11 | | | | | |
| 12 | | | | | |
| Cycles delayed | | n | <b>%</b> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Cycles delayed | | | | | |
| Cycles omitted | | n | <sub>%</sub> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Cycles omitted | | | | | |
| <sup>1</sup> Calculated percentag | ge from t | he total of patien | ts with available data | | |
| | T | able 87 Adhere | ence to Tremelimum | ab in cohort 2 | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Cycles received | | | | | |
| 4 Cycles received | | n | <b>%</b> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| Cycles received | | n | <sub>%</sub> 1 | 95% CI o | f the proportion |
| 0 | | | - | | |
| 1 | | | | | |

Statistical Analysis Plan
Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20




| 3 | | | | | |
|---|---|---|---|---|---|
| 4 | | | | | |
| Cycles delayed | | n | <b>%</b> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Cycles delayed | | | | | |
| Cycles omitted | | n | <sub>%</sub> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Cycles omitted | | | | | |

 $<sup>^{\,1}</sup>$  Calculated percentage from the total of patients with available data

## 1.3.3 Study medication in cohort 3

For the descriptive analysis of the patients, the full analysis set is used (see section 29).

#### Table 88 Adherence to Durvalumab in cohort 3

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|---|---|---|---|---|---|
| Cycles received | | | | | |
| 12 Cycles received | | n | <b>%</b> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| Cycles received | | n | % <sup>1</sup> | 95% CI o | f the proportion |
| 0 | | | | | |
| 1 | | | | | |
| 2 | | | | | |
| 3 | | | | | |
| 4 | | | | | |
| 5 | | | | | |
| 6 | | | | | |
| 7 | | | | | |
| 8 | | | | | |
| 9 | | | | | |

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT Nº: 2016-002858-20




| 10 | | | | | |
|---|---|---|---|---|---|
| 11 | | | | | |
| 12 | | | | | |
| Cycles delayed | | n | <sub>%</sub> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Cycles delayed | | | | | |
| Cycles omitted | | n | <sub>%</sub> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Cycles omitted | | | | | |

 $<sup>^{</sup>m 1}$  Calculated percentage from the total of patients with available data

#### Table 89 Adherence to Tremelimumab in cohort 3

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|---|---|---|---|---|---|
| Cycles received | | | | | |
| 4 Cycles received | | n | % <sup>1</sup> | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| Cycles received | | n | <b>%</b> 1 | 95% CI o | f the proportion |
| 0 | | | | | |
| 1 | | | | | |
| 2 | | | | | |
| 3 | | | | | |
| 4 | | | | | |
| Cycles delayed | | n | % <sup>1</sup> | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Cycles delayed | | | | | |
| Cycles omitted | | n | <b>%</b> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |

EudraCT Nº: 2016-002858-20


#### **Cycles omitted**

 $\overline{\phantom{a}^1}$  Calculated percentage from the total of patients with available data



## 1.3.4 Study medication in cohort 4

For the descriptive analysis of the patients, the full analysis set is used (see section 29).

#### Table 90 Adherence to Durvalumab in cohort 4

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|---|---|---|---|---|---|
| Cycles received | | | | | |
| 12 Cycles received | | n | <b>%</b> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| Cycles received | | n | <b>%</b> 1 | 95% CI o | f the proportion |
| 0 | | | | | |
| 1 | | | | | |
| 2 | | | | | |
| 3 | | | | | |
| 4 | | | | | |
| 5 | | | | | |
| 6 | | | | | |
| 7 | | | | | |
| 8 | | | | | |
| 9 | | | | | |
| 10 | | | | | |
| 11 | | | | | |
| 12 | | | | | |
| Cycles delayed | | n | <b>%</b> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Cycles delayed | | | | | |
| Cycles omitted | | n | % <sup>1</sup> | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |

EudraCT Nº: 2016-002858-20






#### Table 91 Adherence to Tremelimumab in cohort 4

| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|---|---|---|---|---|---|
| Cycles received | | | | | |
| 4 Cycles received | | n | <sub>%</sub> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| Cycles received | | n | <b>%</b> 1 | 95% CI o | f the proportion |
| 0 | | | | | |
| 1 | | | | | |
| 2 | | | | | |
| 3 | | | | | |
| 4 | | | | | |
| Cycles delayed | | n | <sub>%</sub> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Cycles delayed | | | | | |
| Cycles omitted | | n | <sub>%</sub> 1 | 95% CI o | f the proportion |
| Yes | | | | | |
| No | | | | | |
| | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
| Cycles omitted | | | | | |

 $<sup>^{\,1}</sup>$  Calculated percentage from the total of patients with available data



Statistical Analysis Plan
Drug Substance DURVALUMAB/TREMELIMUMAB
Study Number ESR 15-11561-DUNE
EudraCT Nº: 2016-002858-20




#### 2 EFFICACY ANALYSES

All efficacy analyses will be based primarily on the Full Analysis Set and secondarily on the Per Protocol Analysis Set.

#### 2.1 PRIMARY EFFICACY ANALYSES

The analysis of clinical benefit rate and overall survival rate will be performed independently for each study cohort when the last patient included in the corresponding cohort of the study will arrived to 9 months after inclusion in the study or have progressed. According to the protocol, the primary objective of the study will be based on the investigator assessment. 9-months clinical benefit rate (CBR) by Response Evaluation Criteria In Solid Tumors (RECIST version 1.1), which is defined as the percentage of patients achieving complete response (CR), partial response (PR), or stable disease (SD) at month 9 after durvalumab plus tremelimumab was started.

#### 2.1.1 Primary efficacy analyses in the Full Analysis Set

The primary endpoint for cohort 1, 2 and 3 is the CBR, nevertheless the result for all the cohorts will be shown below:

Table 92 Clinical benefit rate (investigator assessment) at 9 months in the Full Analysis Set

| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|---|---|---|---|---|---|
| CBR at 9 months | n (%, Cl 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, Cl 95%) |
| Yes (CR, PR, SD) | | | | | |
| No (PD) | | | | | |
| Total | n (100%) | n (100%) | n (100%) | n (100%) | n (100%) |

The primary endpoint for cohort 4 is 9-months overall survival rate, which is defined as the percentage of patients alive at 9 months after durvalumab plus tremelimumab was started, nevertheless the result for all the cohorts will be shown in the following table.

Table 93 Overall survival rate at 9 months in the Full Analysis Set

Study Number ESR 15-11561-DUN EudraCT №: 2016-002858-20




| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|---|---|---|---|---|---|
| Overall survival rate at 9 months | n (%, CI 95%) | n (%, Cl 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, Cl 95%) |
| Alive | | | | | |
| Death | | | | | |
| Total | n (100%) | n (100%) | n (100%) | n (100%) | n (100%) |

Concordance between investigator assessment and independent central radiology review will be analyzed using Cohen's Kappa. Although no significant differences are expected, a sensitivity analysis for the primary efficacy analysis will be performed using as response variable independent central radiology assessment.

Table 94 Agreement in CBR by Cohen's kappa coefficient in the Full Analysis Set

| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|---|---|---|---|---|---|
| CBR at 9 months | Kappa k | Kappa k | Kappa k | Kappa k | Kappa k |
| Investigator assessment vs. | | | | | |
| Independent review | | | | | |

9-months clinical benefit rate (CBR) by Response Evaluation Criteria In Solid Tumors (RECIST version 1.1), according to independent central radiology.

Table 95 Clinical benefit rate (independent central radiology ) at 9 months in the Full Analysis Set

| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|---|---|---|---|---|---|
| CBR at 9 months | n (%, CI 95%) | n (%, Cl 95%) | n (%, CI 95%) | n (%, Cl 95%) | n (%, Cl 95%) |
| Yes (CR, PR, SD) | | | | | |
| No (PD) | | | | | |
| Total | n (100%) | n (100%) | n (100%) | n (100%) | n (100%) |
EudraCT Nº: 2016-002858-20




# 2.1.2 Primary efficacy analyses in the Per Protocol Analysis Set

The primary endpoint for cohort 1, 2 and 3 is the CBR, nevertheless the result for all the cohorts will be shown below:

Table 96 Clinical benefit rate (investigator assessment) at 9 months in the Per Protocol Analysis Set

| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|---|---|---|---|---|---|
| CBR at 9 months | n (%, CI 95%) | n (%, Cl 95%) | n (%, Cl 95%) | n (%, Cl 95%) | n (%, Cl 95%) |
| Yes (CR, PR, SD) | | | | | |
| No (PD) | | | | | |
| Total | n (100%) | n (100%) | n (100%) | n (100%) | n (100%) |

The primary endpoint for cohort 4 is 9-months overall survival rate, which is defined as the percentage of patients alive at 9 months after durvalumab plus tremelimumab was started, nevertheless the result for all the cohorts will be shown in the following table.

Table 97 Overall survival rate at 9 months in the Per Protocol Analysis Set

| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|---|---|---|---|---|---|
| Overall survival rate at 9 months | n (%, CI 95%) | n (%, Cl 95%) | n (%, Cl 95%) | n (%, CI 95%) | n (%, CI 95%) |
| Alive | | | | | |
| Death | | | | | |
| Total | n (100%) | n (100%) | n (100%) | n (100%) | n (100%) |

Concordance between investigator assessment and independent central radiology review will be analyzed using Cohen's Kappa. Although no significant differences are expected, a sensitivity analysis for the primary efficacy analysis will be performed using as response variable independent

Version Number: 1.1 dated on 30/NOV/2017 central radiology assessment.



## Table 98 Agreement in CBR by Cohen's kappa coefficient in the Per Protocol Analysis Set

| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|---|---|---|---|---|---|
| CBR at 9 months | Kappa k | Kappa k | Kappa k | Kappa k | Kappa k |
| Investigator assessment vs. Independent review | | | | | |

9-months clinical benefit rate (CBR) by Response Evaluation Criteria In Solid Tumors (RECIST version 1.1), according to independent central radiology.

Table 99 Clinical benefit rate (independent central radiology ) at 9 months in the Per Protocol Analysis Set

| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|---|---|---|---|---|---|
| CBR at 9 months | n (%, Cl 95%) | n (%, Cl 95%) | n (%, Cl 95%) | n (%, Cl 95%) | n (%, Cl 95%) |
| Yes (CR, PR, SD) | | | | | |
| No (PD) | | | | | |
| Total | n (100%) | n (100%) | n (100%) | n (100%) | n (100%) |




### 2.2 SECONDARY EFFICACY ANALYSES

The analysis of clinical benefit rate and overall survival rate will be performed independently for each study cohort when the last patient included in the corresponding cohort of the study will arrived to 9 months after inclusion in the study or have progressed. According to the protocol, the secondary objectives of the study will be based on the investigator assessment. 9-months clinical benefit rate (CBR) by Immune-related Response Evaluation Criteria In Solid Tumors (irRECIST), is defined as the percentage of patients achieving complete response (CR), partial response (PR), or stable disease (SD) at month 9 after durvalumab plus tremelimumab was started.

#### 2.2.1 Overall response rate (ORR)

The Overall response rate (ORR) by irRECIST and the duration of the response is shown in the following tables for the Full Analysis Set:

#### Table 100 ORR in the Full Analysis Set

| Cohort 1<br>n (%, CI 95%) | Cohort 2<br>n (%, CI 95%) | Cohort 3<br>n (%, CI 95%) | Cohort 4<br>n (%, Cl 95%) | Total<br>n (%, CI 95%) |
|---|---|---|---|---|
| n (%, CI 95%) | n (%, Cl 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, CI 95%) |
| | | | | . , , |
| n (100%) | n (100%) | n (100%) | n (100%) | n (100%) |
| n (100%) | n (100%) | n (100%) | n (100%) | n (100%) |

EudraCT Nº: 2016-002858-20




## Table 101 Duration of the response in the Full Analysis Set

| Duration of the response (months) | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|---|---|---|---|---|---|
| Cohort 1 | | | | | |
| Cohort 2 | | | | | |
| Cohort 3 | | | | | |
| Cohort 4 | | | | | |
| Total | | | | | |

The Overall response rate (ORR) by irRECIST and the duration of the response is shown in the following table for the Per Protocol Analysis Set:

## Table 102 ORR in the Per Protocol Analysis Set

| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|---|---|---|---|---|---|
| ORR | n (%, Cl 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, Cl 95%) |
| CR | | | | | |
| PR | | | | | |
| SD | | | | | |
| PD | | | | | |
| Total | n (100%) | n (100%) | n (100%) | n (100%) | n (100%) |
| CR or PR | | | | | |
| SD or PD | | | | | |
| Total | n (100%) | n (100%) | n (100%) | n (100%) | n (100%) |

EudraCT Nº: 2016-002858-20




### Table 103 Duration of the response in the Per Protocol Analysis Set

| Duration of the response (months) | n | Mean (SD) | Median (IQR) | Min-Max | 95% CI of the mean |
|---|---|---|---|---|---|
| Cohort 1 | | | | | |
| Cohort 2 | | | | | |
| Cohort 3 | | | | | |
| Cohort 4 | | | | | |
| Total | | | | | |

# 2.2.2 Response status at 6 and 12 months

The response status according to irRECIST at 6 and 12 months after start of study treatment is shown in the following tables for the Full Analysis Set:

Table 104 Response status at 6 months in the Full Analysis Set

| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|---|---|---|---|---|---|
| Response at 6 months | n (%, Cl 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, Cl 95%) |
| CR | | | | | |
| PR | | | | | |
| SD | | | | | |
| PD | | | | | |
| Total | n (100%) | n (100%) | n (100%) | n (100%) | n (100%) |
| CR or PR | | | | | |
| SD or PD | | | | | |

EudraCT Nº: 2016-002858-20


Total

n (100%)

GETNE
Grupo Español de Tumores
Neuroendocrinos

| Neuroendocrinos | | |
|-----------------|----------|----------|
| n (100%) | n (100%) | n (100%) |

### Table 105 Response status at 12 months in the Full Analysis Set

n (100%)

| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|---|---|---|---|---|---|
| Response at 12 months | n (%, Cl 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, CI 95%) |
| CR | | | | | |
| PR | | | | | |
| SD | | | | | |
| PD | | | | | |
| Total | n (100%) | n (100%) | n (100%) | n (100%) | n (100%) |
| CR or PR | | | | | |
| SD or PD | | | | | |
| Total | n (100%) | n (100%) | n (100%) | n (100%) | n (100%) |

The response status according to irRECIST at 6 and 12 months after start of study treatment is shown in the following tables in the Per Protocol Analysis Set:

# Table 106 Response status at 6 months in the Per Protocol Analysis Set

| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|---|---|---|---|---|---|
| Response at 6 months | n (%, CI 95%) | n (%, Cl 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, Cl 95%) |
| CR | | | | | |
| PR | | | | | |

GETNE
Grupo Español de Tumores
Neuroendocrinos

| SD | | | | | |
|---|---|---|---|---|---|
| PD | | | | | |
| Total | n (100%) | n (100%) | n (100%) | n (100%) | n (100%) |
| CR or PR | | | | | |
| SD or PD | | | | | |
| Total | n (100%) | n (100%) | n (100%) | n (100%) | n (100%) |
| | Table 107 Response s | status at 12 months | in the Per Protocol A | nalysis Set | |
| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
| Response at 12 months | n (%, Cl 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, Cl 95%) |
| CR | | | | | |
| PR | | | | | |
| SD | | | | | |
| PD | | | | | |
| Total | n (100%) | n (100%) | n (100%) | n (100%) | n (100%) |
| CR or PR | | | | | |
| SD or PD | | | | | |
| Total | n (100%) | n (100%) | n (100%) | n (100%) | n (100%) |

EudraCT Nº: 2016-002858-20




#### **Progression Free Survival (PFS)** 2.2.3

The median progression-free survival time (PFS) according to irRECIST, along with PFS at 6 and 12 months is shown in the following tables for the Full Analysis Set:

Table 108 Progression Free Survival in the Full Analysis Set

| | | Number of PD | N of patients at risk | | ve progression free<br>urvival | 95% CI of PFS |
|---|---|---|---|---|---|---|
| | Cohort 1 | | | | | |
| | Cohort 2 | | | | | |
| At 6 months | Cohort 3 | | | | | |
| | Cohort 4 | | | | | |
| | Total | | | | | |
| | Cohort 1 | | | | | |
| | Cohort 2 | | | | | |
| At 12 months | Cohort 3 | | | | | |
| | Cohort 4 | | | | | |
| | Total | | | | | |
| | | N (%) of PD | Median (months) | Min-Max | Standard error | 95% CI of the median |
| | Cohort 1 | | | | | |
| | Cohort 2 | | | | | |
| Progression Free<br>Survival | Cohort 3 | | | | | |
| , a. 1. vai | Cohort 4 | | | | | |
| | Total | | | | | |



Figure 1. Progression Free Survival (Full Analysis Set)








The median progression-free survival time (PFS) according to irRECIST, along with PFS at 6 and 12 months is shown in the following tables for the Per-Protocol Analysis Set:

### Table 109 Progression Free Survival in the Per-Protocol Analysis Set

| | | Number of PD | N of patients at risk | | ve progression free<br>urvival | 95% CI of PFS |
|---|---|---|---|---|---|---|
| | Cohort 1 | | | | | |
| | Cohort 2 | | | | | |
| At 6 months | Cohort 3 | | | | | |
| | Cohort 4 | | | | | |
| | Total | | | | | |
| | Cohort 1 | | | | | |
| | Cohort 2 | | | | | |
| At 12 months | Cohort 3 | | | | | |
| | Cohort 4 | | | | | |
| | Total | | | | | |
| | | N (%) of PD | Median (months) | Min-Max | Standard error | 95% CI of the median |
| | Cohort 1 | | | | | |
| | Cohort 2 | | | | | |
| Progression Free<br>Survival | Cohort 3 | | | | | |
| | Cohort 4 | | | | | |
| | Total | | | | | |



Figure 2. Progression Free Survival (Per-Protocol Analysis Set)








# 2.2.4 Overall Survival (OS)

The median overall survival time (OS), along with OS at 6 and 12 months is shown in the following tables for the Full Analysis Set:

### Table 110 Overall Survival in the Full Analysis Set

| | | Number of exitus | N of patients at risk | % of cumulati | ve overall survival | 95% CI of OS |
|---|---|---|---|---|---|---|
| | Cohort 1 | | | | | |
| | Cohort 2 | | | | | |
| At 6 months | Cohort 3 | | | | | |
| | Cohort 4 | | | | | |
| | Total | | | | | |
| | Cohort 1 | | | | | |
| | Cohort 2 | | | | | |
| At 12 months | Cohort 3 | | | | | |
| | Cohort 4 | | | | | |
| | Total | | | | | |
| | | N (%) of exitus | Median (months) | Min-Max | Standard error | 95% CI of the median |
| | Cohort 1 | | | | | |
| | Cohort 2 | | | | | |
| Overall Survival | Cohort 3 | | | | | |
| | Cohort 4 | | | | | |
| | Total | | | | | |



Figure 3. Overall Survival (Full Analysis Set)



| Version Number: 1.1 dated on 30/NOV/2017 | Neuroendocrinos |
|---|---|
| The state of the s | |

GETNE
Grupo Español de Tumores
Neuroendocrinos


The median overall survival time (OS), along with OS at 6 and 12 months is shown in the following tables for the Per-Protocol Analysis Set:

## Table 111 Overall Survival in the Per-Protocol Analysis Set

| | | Number of exitus | N of patients at risk | % of cumulati | ve overall survival | 95% CI of OS |
|---|---|---|---|---|---|---|
| | Cohort 1 | | | | | |
| | Cohort 2 | | | | | |
| At 6 months | Cohort 3 | | | | | |
| | Cohort 4 | | | | | |
| | Total | | | | | |
| | Cohort 1 | | | | | |
| | Cohort 2 | | | | | |
| At 12 months | Cohort 3 | | | | | |
| | Cohort 4 | | | | | |
| | Total | | | | | |
| | | N (%) of exitus | Median (months) | Min-Max | Standard error | 95% CI of the median |
| | Cohort 1 | | | | | |
| | Cohort 2 | | | | | |
| Overall Survival | Cohort 3 | | | | | |
| | Cohort 4 | | | | | |
| | Total | | | | | |

EudraCT Nº: 2016-002858-20




# Figure 4. Progression Free Survival (Per-Protocol Analysis Set)

| The purposition of the foreign or with records. |
|-------------------------------------------------|




## **3** SAFETY ANALYSES

The aim of this section is to assess the safety profile of durvalumab and tremelimumab in subjects with advanced neuroendocrine neoplasms.

# 3.1 MOST FREQUENT TOXICITIES

In the following tables, the most frequent toxicities, those which presented a frequency>10% will be anlayzed in overall and by cohort.

Table 112 Most frequent toxicities in overall

| | | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|---|---|---|---|---|---|---|
| | | n (%, 95% CI) | n (%, 95% CI) | n (%, 95% CI) | n (%, 95% CI) | n (%, 95% CI) |
| | Yes | | | | | |
| Toxicity 1 | No | | | | | |
| | Total | | | | | |
| | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| Grade toxicity 1 | Grade 3 | | | | | |
| • | Grade 4 | | | | | |
| | Total | | | | | |
| | Yes | | | | | |
| Toxicity 2 | No | | | | | |
| | Total | | | | | |
| | Grade 1 | | | | | |
| Crada tavisitu 2 | Grade 2 | | | | | |
| Grade toxicity 2 | Grade 3 | | | | | |
| | Grade 4 | | | | | |

EudraCT Nº: 2016-002858-20




| <br>Total |
|-------------|
| Yes |
| <br>No |
| Total |
| Grade 1 |
| Grade 2 |
| <br>Grade 3 |
| Grade 4 |
| Total |

# **3.2 TOXICITIES GRADE≥3**

In the following table, the number and relative frequencies of patients with at least one grade ≥3 toxicity are summarised:

**Table 113 Toxicities grade ≥3 during follow-up** 

| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|---|---|---|---|---|---|
| Toxicities grade 3 | n (%, Cl 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, CI 95%) |
| Yes | | | | | |
| No | | | | | |
| Total | n (100%) | n (100%) | n (100%) | n (100%) | n (100%) |

In the following table, every toxicity grade ≥3 will be summarised, separately in each one of the 4 cohorts and in overall.

Table 114 Every toxicity grade ≥3 in overall and by cohort

| Cohort 1 Cohort 2 Cohort 3 Cohort 4 Total |
|-------------------------------------------|
|-------------------------------------------|

GETNE
Grupo Español de Tumores
Neuroendocrinos


| Toxicities | n (%, CI 95%) | n (%, Cl 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, Cl 95%) |
|---|---|---|---|---|---|
| Toxicity 1 G≥3 | | | | | |
| Toxicity 2 G≥3 | | | | | |
| Toxicity 3 G≥3 | | | | | |
| Toxicity 4 G≥3 | | | | | |
| Toxicity 5 G≥3 | | | | | |
| Toxicity 6 G≥3 | | | | | |
| Toxicity 7 G≥3 | | | | | |

In the following table, details of every toxicity grade ≥3 will be summarised:

# Table 115 Details of every toxicity grade ≥3 by patient

| Patient number | Hospital | Cohort | Toxicity | Grade |
|----------------|----------|--------|----------|-------|




# 3.3 EVERY TOXICITY

In the following table, the number and relative frequencies of patients with at least one toxicity are summarised:

Table 116 Patients with at least one toxicity during follow-up

| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|---|---|---|---|---|---|
| At least one toxicity | n (%, CI 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, Cl 95%) |
| Yes | | | | | |
| No | | | | | |
| Total | n (100%) | n (100%) | n (100%) | n (100%) | n (100%) |

In the following table, every toxicity grade ≥3 will be summarised, separately in each one of the 4 cohorts and in overall.

Table 117 Every toxicity grade ≥3 in overall and by cohort

| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total |
|---|---|---|---|---|---|
| Toxicities | n (%, CI 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, CI 95%) | n (%, CI 95%) |
| Toxicity 1 G1 | | | | | |
| Toxicity 1 G2 | | | | | |
| Toxicity 1 G3 | | | | | |
| Toxicity 1 G4 | | | | | |
| Toxicity 2 G1 | | | | | |
| Toxicity 2 G2 | | | | | |
| Toxicity 2 G3 | | | | | |
| Toxicity 2 G4 | | | | | |
| Toxicity 3 G1 | | | | | |

EudraCT Nº: 2016-002858-20




| Toxicity 3 G2 |
|-----------------------|
| Toxicity 3 G <i>3</i> |
| Toxicity 3 G4 |

#### 4 EXPLORATORY ANALYSES

The aims of this section are:

- To evaluate biochemical response (changes in CgA and NSE levels) and its association with response rate and progression-free survival.
- To assess whether baseline tumor and blood biomarkers may be predictive of response to durvalumab and tremelimumab therapy.
- To explore additional hypotheses related to biomarkers and relationship to durvalumab and tremelimumab efficacy and/or toxicity and neuroendocrine tumors evolution that may arise from internal or external research activities.

# 4.1 LOGISTIC REGRESSION: PREDICTOR FACTORS OF RESPONSE (CBR AT 9 MONTHS) IN EACH COHORT

A multivariate analysis will be carried out using the Logistic Regression model in order to determine predictor factors for response (CBR at 9 months) in each cohort. Firstly univariate analysis are carried out separately for each one of the possible predictor factors to decide which variables are entered in the multivariate models; only those with a statistical association with the dependent variable would be selected. Backward elimination stepwise process would be used to select the model. In the first step all possible predictors are entered in the model and in each step, the variable that is least significant (that is, the one with the largest P value) is removed and the model is refitted. Each subsequent step removed the least significant variable in the model until all remaining variables have individual P values smaller than 0.05.

Table 118 Univariate Logistic Regression for Response (CBR at 9 months) in cohort 1 (Full Analysis Set)

| | p-value (variable) | OR | CI 95% of OR | N | p-value (categories) |
|----------|--------------------|----|--------------|---|----------------------|
| Factor 1 | Category 1 | | | | |
| ractor 1 | Category 2 | | | | |

Statistical Analysis Plan

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT №: 2016-002858-20




| Factor 2 | Category 1 |
|----------|------------|
| FACTOR 2 | Category 2 |
| Factor 3 | Category 1 |
| ractor 5 | Category 2 |
| Factor 4 | Category 1 |
| ractor 4 | Category 2 |
| | Category 1 |
| | Category 2 |

## Table 119 Final multivariate Logistic Regression for Response (CBR at 9 months) in cohort 1 (Full Analysis Set)

| p-va | lue (variable) | OR | CI 95% of OR | N | p-value (categories) |
|----------|----------------|----|--------------|---|----------------------|
| Factor 1 | Category 1 | | | | |
| Factor 1 | Category 2 | | | | |
| Factor 2 | Category 1 | | | | |
| Factor 2 | Category 2 | | | | |
| | Category 1 | | | | |
| ••• | Category 2 | | | | |

# Table 120 Univariate Logistic Regression for Response (CBR at 9 months) in cohort 2 (Full Analysis Set)

| | p-value (variable) | OR | CI 95% of OR | N | p-value (categories) |
|----------|--------------------|----|--------------|---|----------------------|
| Factor 1 | Category 1 | | | | |
| racioi 1 | Category 2 | | | | |

Statistical Analysis Plan

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT №: 2016-002858-20




| Category 1 |
|------------|
| Category 2 |
| Category 1 |
| Category 2 |
| Category 1 |
| Category 2 |
| Category 1 |
| Category 2 |

## Table 121 Final multivariate Logistic Regression for Response (CBR at 9 months) in cohort 2 (Full Analysis Set)

| p-v | alue (variable) | OR | CI 95% of OR | N | p-value (categories) |
|----------|-----------------|----|--------------|---|----------------------|
| Fastor 1 | Category 1 | | | | |
| Factor 1 | Category 2 | | | | |
| Footow 2 | Category 1 | | | | |
| Factor 2 | Category 2 | | | | |
| | Category 1 | | | | |
| ••• | Category 2 | | | | |

# Table 122 Univariate Logistic Regression for Response (CBR at 9 months) in cohort 3 (Full Analysis Set)

| p-va | llue (variable) | OR | CI 95% of OR | N | p-value (categories) |
|----------|-----------------|----|--------------|---|----------------------|
| Footow 1 | Category 1 | | | | |
| Factor 1 | Category 2 | | | | |
| Factor 2 | Category 1 | | | | |

Statistical Analysis Plan

Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT №: 2016-002858-20




| | Category 2 |
|-----|------------|
| | Category 1 |
| ••• | Category 2 |

| p-v | alue (variable) | OR | CI 95% of OR | N | p-value (categories) |
|----------|-----------------|----|--------------|---|----------------------|
| Factor 1 | Category 1 | | | | |
| Factor 1 | Category 2 | | | | |
| Factor 2 | Category 1 | | | | |
| Factor 2 | Category 2 | | | | |
| | Category 1 | | | | |
| ••• | Category 2 | | | | |

# Table 124 Univariate Logistic Regression for Response (CBR at 9 months) in cohort 4 (Full Analysis Set)

| p | -value (variable) | OR | CI 95% of OR | N | p-value (categories) |
|----------|-------------------|----|--------------|---|----------------------|
| Factor 1 | Category 1 | | | | |
| Factor 1 | Category 2 | | | | |
| Factor 2 | Category 1 | | | | |
| Factor 2 | Category 2 | | | | |

Statistical Analysis Plan
Drug Substance DURVALUMAB/TREMELIMUMAB

Study Number ESR 15-11561-DUNE EudraCT №: 2016-002858-20




| Factor 3 | Category 1 |
|----------|------------|
| ractor 5 | Category 2 |
| Factor 4 | Category 1 |
| ractor 4 | Category 2 |
| | Category 1 |
| ••• | Category 2 |

### Table 125 Final multivariate Logistic Regression for Response (CBR at 9 months) in cohort 4 (Full Analysis Set)

| p-v | alue (variable) | OR | CI 95% of OR | N | p-value (categories) |
|----------|-----------------|----|--------------|---|----------------------|
| Factor 1 | Category 1 | | | | |
| ractor 1 | Category 2 | | | | |
| Footow 2 | Category 1 | | | | |
| Factor 2 | Category 2 | | | | |
| | Category 1 | | | | |
| ••• | Category 2 | | | | |

### 4.2 COX REGRESSION: PREDICTOR FACTORS OF SURVIVAL IN EACH COHORT

# 4.2.1 Cox Regression: predictor factors of PFS in each cohort

A multivariate analysis will be carried out using the Cox Regression model in order to determine predictor fators for PFS *in each cohort*. Firstly univariate analysis are carried out separately for each one of the possible predictor factors to decide which variables are entered in the multivariate models; only those with a statistical association with the dependent variable would be selected. Backward elimination stepwise process would be used to select the model. In the first step all possible predictors are entered in the model and in each step, the variable that is least significant (that is, the one with the largest P value) is removed and the model is refitted. Each subsequent step removed the least significant variable in the model until

EudraCT Nº: 2016-002858-20


all remaining variables have individual P values smaller than 0.05.



# Table 126 Univariate Cox Regression for PFS in cohort 1 (Full Analysis Set)

| | | HR | CI 95% of HR | p-value | n |
|---|---|---|---|---|---|
| ·1 | Category 1 | | | | |
| actor 1 | Category 2 | | | | |
| actor 2 | Category 1 | | | | |
| actor 2 | Category 2 | | | | |
| actor 3 | Category 1 | | | | |
| actor 5 | Category 2 | | | | |
| actor 4 | Category 1 | | | | |
| actor 4 | Category 2 | | | | |
| | Category 1 | | | | |
| •• | Category 2 | | | | |
| | Table 127 | Final multivariate Cox Reg | ression for PFS in cohort 1 (Fu | ıll Analysis Set) | |
| | | HR | CI 95% of HR | p-value | n |
| · 1 | Category 1 | | | | |
| actor 1 | Category 2 | | | | |
| anton 3 | Category 1 | | | | |
| actor 2 | Category 2 | | | | |
| | Category 1 | | | | |



| version number: 1 | | | | | |
|---|---|---|---|---|---|
| | | HR | CI 95% of HR | p-value | n |
| Factor 1 | Category 1 | | | | |
| | Category 2 | | | | |
| | Category 1 | | | | |
| Factor 2 | Category 2 | | | | |
| Footow 2 | Category 1 | | | | |
| Factor 3 | Category 2 | | | | |
| 5t 4 | Category 1 | | | | |
| Factor 4 | Category 2 | | | | |
| | Category 1 | | | | |
| ••• | Category 2 | | | | |
| | category 2 | | | | |
| | | nal multivariate Cox Reg | ression for PFS in cohort 2 (Fu | II Analysis Set) | |
| | | nal multivariate Cox Regi | ression for PFS in cohort 2 (Fu | ll Analysis Set) | n |
| | | | | | n |
| Factor 1 | Table 129 Fi | | | | n |
| | Table 129 File | | | | n |
| | Category 1 Category 2 | | | | n |
| | Category 1 Category 2 Category 1 | | | | n |
| Factor 1 Factor 2 | Category 1 Category 2 Category 1 Category 2 | | | | n |
| Factor 2 | Category 1 Category 2 Category 1 Category 2 Category 2 Category 2 Category 1 | | | | n |
| Factor 2 | Category 1 Category 2 Category 2 Category 2 Category 2 Category 1 Category 2 Category 1 | HR | | p-value | n |

EudraCT Nº: 2016-002858-20



| Factor 1 | Category 1 | | | | |
|---|---|---|---|---|---|
| ractor 1 | Category 2 | | | | |
| Factor 2 | Category 1 | | | | |
| ractor 2 | Category 2 | | | | |
| Factor 3 | Category 1 | | | | |
| | Category 2 | | | | |
| Factor 4 | Category 1 | | | | |
| | Category 2 | | | | |
| | Category 1 | | | | |
| ••• | Category 2 | | | | |
| | Table 131 F | Final multivariate Cox Reg | ression for PFS in cohort 3 (Fu | ıll Analysis Set) | |
| | Table 131 F | Final multivariate Cox Regi | ression for PFS in cohort 3 (Fu<br>CI 95% of HR | ull Analysis Set) p-value | n |
| Castor 1 | Table 131 F | | | | n |
| actor 1 | | | | | n |
| | Category 1 | | | | n |
| | Category 1 Category 2 | | | | n |
| | Category 1 Category 2 Category 1 | | | | n |
| Factor 1 Factor 2 | Category 1 Category 2 Category 1 Category 2 | | | | n |
| Factor 2 | Category 1 Category 2 Category 1 Category 2 Category 1 Category 2 | HR | | p-value | n |
| Factor 2 | Category 1 Category 2 Category 1 Category 2 Category 1 Category 2 | HR | CI 95% of HR | p-value | n |
| Factor 2 | Category 1 Category 2 Category 1 Category 2 Category 1 Category 2 | HR<br>32 Univariate Cox Regress | CI 95% of HR ion for PFS in cohort 4 (Full A | p-value<br>nalysis Set) | |



| Factor 2 | Category 1 | | | | |
|---|---|---|---|---|---|
| ractor 2 | Category 2 | | | | |
| Factor 3 | Category 1 | | | | |
| | Category 2 | | | | |
| Factor 4 | Category 1 | | | | |
| | Category 2 | | | | |
| | Category 1 | | | | |
| ••• | Category 2 | | | | |
| ••• | | Final multivariate Cox Reg | ression for PFS in cohort 4 (Fo | ıll Analysis Set) | |
| ··· | | Final multivariate Cox Reg<br>HR | ression for PFS in cohort 4 (Fo | ull Analysis Set) p-value | n |
| | | | | | n |
| | Table 133 | | | | n |
| Factor 1 | Table 133 | | | | n |
| Factor 1 | Category 1 Category 2 | | | | n |
| Factor 1 | Category 1 Category 2 Category 1 | | | | n |

EudraC1 Nº: 2016-002858-20




# 4.2.2 Cox Regression: predictor factors of OS in each cohort

A multivariate analysis will be carried out using the Cox Regression model in order to determine predictor fators for OS *in each cohort*. Firstly univariate analysis are carried out separately for each one of the possible predictor factors to decide which variables are entered in the multivariate models; only those with a statistical association with the dependent variable would be selected. Backward elimination stepwise process would be used to select the model. In the first step all possible predictors are entered in the model and in each step, the variable that is least significant (that is, the one with the largest P value) is removed and the model is refitted. Each subsequent step removed the least significant variable in the model until all remaining variables have individual P values smaller than 0.05.

Table 134 Univariate Cox Regression for OS in cohort 1 (Full Analysis Set)

| | | HR | CI 95% of HR | p-value | n |
|---|---|---|---|---|---|
| Fastau 1 | Category 1 | | | | |
| Factor 1 | Category 2 | | | | |
| Factor 2 | Category 1 | | | | |
| Factor 2 | Category 2 | | | | |
| Footow 2 | Category 1 | | | | |
| Factor 3 | Category 2 | | | | |
| | Category 1 | | | | |
| Factor 4 | Category 2 | | | | |
| | Category 1 | | | | |
| •• | Category 2 | | | | |
| | Table 135 | Final multivariate Cox Reg | ression for OS in cohort 1 (Fu | ll Analysis Set) | |
| | | HR | CI 95% of HR | p-value | n |
| Fastau 1 | Category 1 | | | | |
| Factor 1 | Category 2 | | | | |

EudraCT Nº: 2016-002858-20




| Factor 2 | Category 1 |
|----------|------------|
| ractor 2 | Category 2 |
| | Category 1 |
| ··· | Category 2 |

# Table 136 Univariate Cox Regression for OS in cohort 2 (Full Analysis Set)

| | | HR | CI 95% of HR | p-value | n |
|---|---|---|---|---|---|
| Factor 1 | Category 1 | | | | |
| ractor 1 | Category 2 | | | | |
| Factor 2 | Category 1 | | | | |
| racioi Z | Category 2 | | | | |
| Factor 3 | Category 1 | | | | |
| ractor 5 | Category 2 | | | | |
| Factor 4 | Category 1 | | | | |
| Factor 4 | Category 2 | | | | |
| | Category 1 | | | | |
| ••• | Category 2 | | | | |
| | Table 137 | ' Final multivariate Cox Reg | ression for OS in cohort 2 (Fu | ll Analysis Set) | |
| | | HR | CI 95% of HR | p-value | n |
| Footow 1 | Category 1 | | | | |
| Factor 1 | Category 2 | | | | |
| Factor 2 | Category 1 | | | | |

GETNE
Grupo Español de Tumores
Neuroendocrinos

| Version Number: 1 | .1 dated on 30/NOV/2017 | | Neuroendocrinos | | |
|---|---|---|---|---|---|
| | Category 2 | | | | |
| | Category 1 | | | | |
| •• | Category 2 | | | | |
| | Table | 138 Univariate Cox Regress | sion for OS in cohort 3 (Full A | nalysis Set) | |
| | | HR | CI 95% of HR | p-value | n |
| actor 1 | Category 1 | | | | |
| actor 1 | Category 2 | | | | |
| actor 2 | Category 1 | | | | |
| actor 2 | Category 2 | | | | |
| ostor 2 | Category 1 | | | | |
| actor 3 | Category 2 | | | | |
| actor 4 | Category 1 | | | | |
| actor 4 | Category 2 | | | | |
| | Category 1 | | | | |
| •• | Category 2 | | | | |
| | Table 139 | Final multivariate Cox Reg | ression for OS in cohort 3 (Fu | ll Analysis Set) | |
| | | HR | CI 95% of HR | p-value | n |
| inatou 1 | Category 1 | | | | |
| actor 1 | Category 2 | | | | |
| t 2 | Category 1 | | | | |
| actor 2 | Category 2 | | | | |
| •• | Category 1 | | | | |

Neuroendocrinos


#### Category 2

### Table 140 Univariate Cox Regression for OS in cohort 4 (Full Analysis Set) HR CI 95% of HR p-value n Category 1 Factor 1 Category 2 Category 1 Factor 2 Category 2 Category 1 Factor 3 Category 2 Category 1 Factor 4 Category 2 Category 1 Category 2 Table 141 Final multivariate Cox Regression for OS in cohort 4 (Full Analysis Set) HR CI 95% of HR p-value n Category 1 Factor 1 Category 2 Category 1 Factor 2 Category 2 Category 1 Category 2




### 5 GENERAL CONSIDERATIONS

# 5.1 TIMING OF ANALYSES

Recruitment period will be: 24 months Research Agreement executed: July 2016 Projected IRB/IEC approval: Nov 2016 First Subject In: Dec 2016 50% Enrollment: Dec2017 Last Subject In (100% enrollment): Dec 2018 Last Subject Last Visit: Dec 2019 Clinical Study Report April 2020

End of study is defined as Last Subject Last Visit.

#### 5.2 REPORTING CONVENTIONS

P-values ≥0.001 will be reported to 3 decimal places; p-values less than 0.001 will be reported as "<0.001". The mean, standard deviation, and any other statistics other than quantiles, will be reported to one decimal place greater than the original data. Quantiles, such as median, or minimum and maximum will use the same number of decimal places as the original data. Estimated parameters, not on the same scale as raw observations (e.g. regression coefficients) will be reported to 3 significant figures.

#### 5.3 TECHNICAL DETAILS

This SAP has been based on the PROTOCOL version 3.1 dated on 30/NOV/2017. R software version 3.2.1 will be used for all analysis (or the last version available at the time of the analysis).

Databases, syntax code and any other files used for the analysis will be electronically stored by

Following standard operating practices (SOPs), working practice documents, and applicable regulations and guidelines.




# 6 REFERENCES

- (1) G.J.M.G. van der Heijden et al. Imputation of missing values is superior to complete case analysis and the missing-indicator method in multivariable diagnostic research: A clinical example. Journal of Clinical Epidemiology 59 (2006) 1102e1109
- (2) European Medicines Agency. Guideline on missing data in confirmatory clinical trials. 2010. www.ema.europa.eu/docs/en\_GB/document\_library/Scientific\_guideline/2010/09/WC500096793.pdf.
- (3) Altman D. Missing outcomes in randomized trials: addressing the dilemma. Open Med2009;3(2):e51.
- (4) Little, R. J., y D. Rubin (2002), Statistical analysis with missing data (Sec. Ed.), New York, Wiley.